## The GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

| Title | ÷ | Reporting and Analysis Plan for FDC116114: Implementation of a screening tool for subjects with benign prostatic enlargement/obstruction to identify men ≥50 years presenting in General Practice with other co-morbidities who should be assessed for BPH |
|---|---|---|
| Compound Number | : | Not Applicable |
| <b>Effective Date</b> | : | 20-APR-2017 |

## **Description:**

• The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report (CSR) for Protocol FDC116114. This document contains the RAP Amendment 01.

#### **Author's Name and Functional Area:**

| | PPD | | |
|---|---|---|---|
| Original | Principal Biostatis | stician, Biostatistics, PAREXEL | 17-FEB-2017 |
| | International Emp | ployee of PAREXEL on behalf of GSK | |
| | PPD | | |
| Amendment | Principal Biostatistician, Biostatistics, PAREXEL | | 19-APR-2017 |
| 01 | International Employee of PAREXEL on behalf of GSK | | |

## Approved by:

| Original | | (email approval dated 28-Feb-2017)<br>atistics & Programming, GSK | 28-FEB-2017 |
|---|---|---|---|
| Amendment 01 | PPD Director Sta | (email approval dated 20-APR-2017) atistics & Programming, GSK | 20-APR-2017 |

Copyright 2017 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# **TABLE OF CONTENTS**

| | | | | PAGE |
|---|---|---|---|---|
| 1. | REPC | RTING & | ANALYSIS PLAN SYNOPSIS | 5 |
| 2. | CLIMAN | | KEY PROTOCOL INFORMATION | 10 |
| ۷. | 2.1. | | | |
| | 2.1. | Change | s to the Protocol Defined Statistical Analysis Plan | 10 |
| | | | bjective(s) and Endpoint(s) | |
| | 2.3. | | esign | |
| | 2.4. | Statistic | al Hypotheses | 14 |
| 3. | PLAN | NED ANA | ALYSES | 14 |
| | 3.1. | Interim A | Analyses | 14 |
| | 3.2. | | alyses | |
| 4. | ΔΝΔΙ | VSIS POI | PULATIONS | 15 |
| \lnot. | 4.1. | | Deviations | |
| | 4.1. | 4.1.1. | | |
| | | 4.1.1. | | |
| | | 4.1.2. | Important Protocol Deviations | 15 |
| 5. | | | ONS FOR DATA ANALYSES AND DATA HANDLING | |
| | CONV | /ENTION: | S | 17 |
| 6. | STUD | Y POPUL | ATION ANALYSES | 18 |
| | 6.1. | Overvie | w of Planned Analyses | 18 |
| | 6.2. | Subject | Accountability | 19 |
| | 6.3. | • | Disposition | |
| | 6.4. | | aphic Characteristics | |
| | 6.5. | Medical | Conditions, Surgical Procedures, and Concomitant | |
| | | | ions | |
| | 6.6. | Diagnos | tic Tests and Questionnaires | 22 |
| 7. | PRIM | ARY STA | TISTICAL ANALYSES | 23 |
| | 7.1. | Primary | Efficacy Analyses | <mark>23</mark> |
| | | 7.1.1. | overview or realistical remaining Emodely remails | |
| | | 7.1.2. | Planned Primary Efficacy Statistical Analyses | 24 |
| 8. | SECC | NDARY S | STATISTICAL ANALYSES | 25 |
| | 8.1. | | ary Efficacy Analyses | |
| | | 8.1.1. | Overview of Planned Secondary Efficacy Analyses | |
| | | 8.1.2. | Planned Secondary Efficacy Statistical Analyses | |
| | | • | 8.1.2.1. IPSS Screening Tool | |
| | | | 8.1.2.2. BPH-Related Health Status | |
| | | | 8.1.2.3. BPE/BPO Screening Tool | |
| | 8.2. | Safety A | Analyses | |
| | 0.2. | 8.2.1. | Overview of Planned Analyses | |
| | | 8.2.2. | Adverse Events | |
| | | 8.2.3. | Deaths and Serious Adverse Events | |
| | | 8.2.4. | Adverse Events Leading to Withdrawal From the Study | |
| | | 0.2.7. | and Other Significant Adverse Events | 33 |
| | | | ANA SUIDI SIANINGANI FAMONO EMPINO | |

| | | 8.2.4.1. | Adverse Events Leading to Withdrawal from | |
|---|---|---|---|---|
| | | | the Study | 33 |
| | | | Adverse Events of Special Interest | 33 |
| | | | Sexual and Breast Tier 1 Adverse Events of | |
| | | | Special Interest | 33 |
| | | | Prostate Cancer Adverse Events of Special | 0.4 |
| | | | Interest | 34 |
| | | | Cardiovascular Adverse Events of Special | 24 |
| | | | Interest | 34 |
| | | 0.2.4.0. | Interest | 34 |
| | | | poratory Assessments | |
| | | | A | |
| | | | tal Examinations | |
| | 8.3. | | alyses | |
| | 8.4. | | and / or Biomarker) Analyses | |
| | 8.5. | | narmacodynamic Ánalyses | |
| | | | · | |
| 9. | OTHE | R STATISTICAL ANA | LYSES | 36 |
| 10. | REFE | RENCES | | 37 |
| 4.4 | ٨٥٥٥ | IDIOEO | | 20 |
| 11. | 11.1. | | I Deviation Management and Definitions for Der | 30 |
| | 11.1. | | I Deviation Management and Definitions for Per | 30 |
| | | 11 1 1 Evolucione | from Per Protocol Population | 30 |
| | 11.2. | | Events | |
| | 11.2. | 11 2 1 Protocol De | efined Time & Events | 40<br>40 |
| | 11.3. | | ment Windows | |
| | 11.4. | | ent States and Phases | |
| | 11.5. | • • | splay Standards & Handling Conventions | |
| | | | tment & Sub-group Display Descriptors | |
| | | | efinition & Derivations | |
| | | 11.5.3. Reporting F | Process & Standards | 44 |
| | 11.6. | Appendix 6: Derived | and Transformed Data | 46 |
| | | 11.6.1. General | | |
| | | | ulation | |
| | 11.7. | | re Withdrawals & Handling of Missing Data | |
| | | | Withdrawals | |
| | | 11.7.2. Handling of | f Missing Data | 48 |
| | | | Handling of Missing Dates | |
| | 11.8. | | Handling of Partial Datese Event Time Periods and Special Adverse | 49 |
| | 11.0. | | Event Time Ferious and Special Adverse | 50 |
| | 11.9. | | of Potential Clinical Importance | |
| | 11.5. | | Values | |
| | 11 10 | , | enter Studies | |
| | | | or Handling Centers | |
| | 11.11. | | nation of Covariates, Subgroups & Other Strata | |
| | 11.12. | | e Comparisons & Multiplicity | |
| | | | f Multiple Comparisons & Multiplicity | |

# 2017N326958\_00 FDC116114

## CONFIDENTIAL

| 11.13. | Appendix 13: Model Checking and Diagnostics for Statistical | |
|--------|-------------------------------------------------------------|----|
| | Analyses | 66 |
| 11.14. | Appendix 14: Abbreviations and Trademarks | 67 |
| | 11.14.1. Abbreviations | 67 |
| | 11.14.2. Trademarks | 67 |
| 11.15. | Appendix 15: List of Data Displays | 68 |
| | 11.15.1. Data Display Numbering | |
| | 11.15.2. Study Population Tables | |
| | 11.15.3. Efficacy Tables | |
| | 11.15.4. Efficacy Figures | 73 |
| | 11.15.5. Safety Tables | |
| | 11.15.6. ICH Listings | 75 |
| 11.16. | Appendix 16: Example Mock Shells for Data Displays | |
| | Appendix 17: Amendment 01 Revision | |

# 1. REPORTING & ANALYSIS PLAN SYNOPSIS

| Overview | Key Elements of the RAP |
|---|---|
| Purpose | The purpose of this Reporting and Analysis Plan (RAP) is to describe the planned summaries and statistical analyses to be included in the Clinical Study Report (CSR) for Protocol FDC116114. |
| Protocol | This RAP is based on protocol amendment 02 (Dated: 18/JAN/2016) of study FDC116114 (GSK Document No. :2012N140248_02] and eCRF Version 2.0.1. This document contains the RAP amendment 01. |
| | The aim of the study is to evaluate the utility of the Benign Prostatic Enlargement (BPE)/Benign Prostatic Obstruction (BPO) screening tool in a general practice setting. The results of this screening tool may be used for further investigation. |
| Primary<br>Objective | The primary objective is to assess the utility of a BPE/BPO screening tool in conjunction with serum prostate specific antigen (PSA) in finding men confirmed to have benign prostatic hyperplasia (BPH) on full Urologist assessment of diagnostic test results. |
| Primary<br>Endpoint | • The primary endpoint is the proportion of men that are confirmed to have BPH based on full Urologist assessment of diagnostic test results among men with a positive result on the BPE/BPO screening tool (score ≥3) and serum PSA≥2 ng/mL. |
| Study | No investigational study drug is being administered during this study. |
| Design | This is a non-randomized, interventional study utilizing a questionnaire-based assessment of men in general practice. Men who sign the informed consent form and meet the eligibility criteria will be enrolled and complete the Part I diagnostic tests at the General Practitioners (GP) clinic. If the GP determines that the subject has probable BPH, the subject proceeds to Part II and is scheduled for a Urologist assessment and diagnostic tests to confirm or refute a BPH diagnosis and to assess risk of progression of BPH. |
| | <ul> <li>Approximately 1,500 males ≥50 years presenting to a GP for a reason that is<br/>not related to this study will be screened for probable BPH to yield 500 subjects<br/>being referred to a Urologist.</li> </ul> |
| | The duration of the study will be 1 week (±4 days) and up to 6 weeks to allow for GP and Urologist visit scheduling. |
| Planned | No investigational study drug is being administered during this study. |
| Analyses | • The primary endpoint is defined as the proportion of men confirmed to have BPH based on full Urologist diagnostic testing among men with a positive result on the BPE/BPO screening tool (score ≥3) and serum PSA ≥2 ng/mL. Primary endpoint summaries will be descriptively presented in terms of the calculated proportion, described below in the Primary Analyses Section, and 95% confidence interval on the proportion. Formal hypothesis testing will not be conducted. |

# Overview **Key Elements of the RAP** Secondary endpoints and other measures of interest are defined in terms of proportions for each: probable BPH diagnosis by GP, BPH diagnosis by Urologist, and BPH progression risk by Urologist along with use of 1) BPE/BPO screening tool and 2) International Prostate Symptom Score (IPSS) screening tool. The 95% confidence intervals for these proportions will be presented. Additional summaries, proportions and related 95% confidence intervals, will be generated as outlined above, but in terms of a positive result for both the BPE/BPO and the IPSS screening tools, and separately for either the BPE/BPO or IPSS screening tools. Another secondary endpoint of this study is to assess the level of agreement between the BPE/BPO and the IPSS screening tools for selecting men to investigate for BPH. The number and proportion of subjects with a positive or with a negative response to both the BPE/BPO and IPSS screening tools at screening will be summarized. Agreement of the BPE/BPO and the IPSS screening tools will be assessed using the kappa coefficient. The simple kappa coefficient along with the 95% confidence interval based on the asymptotic standard error will be generated using SAS. The associated null hypothesis is that the two measures (BPE/BPO and IPSS screening tools) are independent, i.e., kappa = 0. The alternative hypothesis is that the agreement of the two measures is better than one would expect by chance. If the 95% confidence interval does not contain the value zero (0), reject the hypothesis that kappa=0 (no agreement) for these data at the 0.05 level of significance. The above defined kappa coefficient will be characterized as proposed by Landis and Koch (Landis, 1977) with <0 indicating no agreement, 0-0.20 as slight, 0.21-0.40 as fair, 0.41-0.60 as moderate, 0.61-0.80 as substantial, and 0.81 – 1 as almost perfect agreement. The proportion of subjects who discontinued from the study before the GP was able to assess the presence of probable BPH will be summarized. The proportion of subjects who withdrew from the study before a Urologist visit, among subjects with a probable GP BPH diagnosis will be summarized. The above described proportions, for both primary and secondary endpoints, will also be summarized by country, and separately by country and center.

| Overview | Key Elements of | the RAP | | |
|---|---|---|---|---|
| Analysis | No investigational study drug is being administered during this study. | | | |
| Populations | Subjects are not randomized or dispensed study treatment. | | | |
| | Population | Definition / Crite | eria | |
| | Screened | Comprised of eligibility. | f all subjects who are | screened for |
| | Screened But No Evaluable | | f all subjects who are s<br>but do not qualify for topulation. | |
| | Evaluable | criteria, includ<br>result (score | | |
| Hypothesis | <ul> <li>The primary endpoint is defined as the proportion of men confirmed to have<br/>BPH based on full Urologist diagnostic testing in men with a positive result on<br/>the BPE/BPO screening tool (score ≥ 3) and a serum PSA ≥ 2 ng/mL. Formal<br/>hypothesis testing will not be conducted in terms of the primary and secondary<br/>endpoint proportions.</li> </ul> | | | |
| Primary<br>Analyses | <ul> <li>The primary endpoint is defined as the proportion of men confirmed to have BPH based on full Urologist diagnostic testing among men with a positive result on the BPE/BPO screening tool (score ≥3) and serum PSA ≥2 ng/mL.</li> <li>Primary endpoint summaries will be descriptively presented in terms of the calculated proportion, described below, and 95% confidence interval on the proportion. Formal hypothesis testing will not be conducted.</li> </ul> Tool Proportion Numerator Denominator | | | |
| | BPE/BPO | BPH diagnosis by Urologist based upon BPE/BPO screening tool result (score≥3) and serum PSA ≥2 ng/mL. | Number of subjects<br>diagnosed with BPH<br>based upon a BPH<br>assessment by<br>Urologist | Number of subjects with a positive result on the BPE/BPO screening tool (score≥3) and serum PSA ≥2 ng/mL and a BPH assessment by Urologist. |

Secondary endpoints and other measures of interest are defined in terms of

Overview

Secondary

**Key Elements of the RAP** 

(score ≥3)

#### Analyses proportions for each: probable BPH diagnosis by GP, BPH diagnosis by Urologist, and BPH progression risk by Urologist along with use of 1) BPE/BPO screening tool and 2) IPSS screening tool. The 95% confidence intervals for these proportions will be presented. Secondary Endpoints: Proportions only in terms of the BPE/BPO tool **Proportion** Tool Numerator **Denominator** BPE/ **BPH Progression Risk** Number of subjects Number of subjects with a BPO by Urologist based diagnosed with BPH positive result on the BPE/BPO upon BPE/BPO screening tool (score ≥3) and progression risk by screening tool result serum PSA ≥2 ng/mL and a Urologist (score ≥3) and serum BPH progression risk PSA ≥2 ng/mL assessment by Urologist BPE/ Probable BPH Number of subjects Number of subjects with a BPO Diagnosis by GP diagnosed with positive result on the BPE/BPO based upon BPE/BPO 'probable BPH' by GP screening tool (score ≥3) and a screening tool result BPH assessment by GP

| Secor | Secondary Endpoints: Proportions only in terms of the IPSS screening tool | | |
|---|---|---|---|
| Tool | Proportion | Numerator | Denominator |
| IPSS | BPH Diagnosis by Urologist based upon IPSS screening result (score ≥8) and serum PSA ≥2 ng/mL | Number of subjects diagnosed with BPH based on a BPH assessment by Urologist. | Number of subjects with a positive result on the IPSS (score ≥8) and serum PSA ≥2 ng/mL and a BPH assessment by Urologist |
| IPSS | BPH Progression Risk<br>by Urologist based<br>upon IPSS screening<br>result (score ≥8) and<br>serum PSA ≥2 ng/mL | Number of subjects<br>diagnosed with BPH<br>progression risk by<br>Urologist | Number of subjects with a positive result on the IPSS (score ≥8) and serum PSA ≥2 ng/mL and a BPH progression risk assessment by Urologist |
| IPSS | Probable BPH Diagnosis by GP based upon IPSS screening result (score ≥8) | Number of subjects diagnosed with 'probable BPH' by GP | Number of subjects with a positive result on the IPSS (score ≥8) and a BPH assessment by GP |

- Additional summaries, proportions and related 95% confidence intervals, will be generated as outlined above, but in terms of a positive result for both the BPE/BPO and the IPSS screening tools and separately for either the BPE/BPO or IPSS screening tools.
- Another secondary endpoint of this study is to assess the level of agreement between the BPE/BPO and IPSS screening tools for selecting men to

| Overview | Key Elements of the RAP |
|---|---|
| | investigate for BPH. The number and proportion of subjects with a positive or with a negative response to both the BPE/BPO and IPSS screening tools at screening will be summarized. |
| | • Agreement of the BPE/BPO and the IPSS screening tools will be assessed using the kappa coefficient. The simple kappa coefficient along with the 95% confidence interval based on the asymptotic standard error will be generated using SAS. The associated null hypothesis is that the two measures (BPE/BPO and IPSS screening tools) are independent, i.e., kappa = 0. The alternative hypothesis is that the agreement of the two measures is better than one would expect by chance. If the 95% confidence interval does not contain the value zero (0), reject the hypothesis that kappa=0 (no agreement) for these data at the 0.05 level of significance. |
| | The above defined kappa coefficient will be characterized as proposed by Landis and Koch (Landis, 1977) with <0 indicating no agreement, 0-0.20 as slight, 0.21-0.40 as fair, 0.41-0.60 as moderate, 0.61-0.80 as substantial, and 0.81 – 1 as almost perfect agreement. |
| | The proportion of subjects who discontinued from the study before the GP was able to assess the presence of probable BPH will be summarized. The proportion of subjects who withdrew from the study before a Urologist visit, among subjects with a probable GP BPH diagnosis will be summarized. |
| | The above described proportions, for both primary and secondary endpoints, will also be summarized by country, and separately by country and center. |

## 2. SUMMARY OF KEY PROTOCOL INFORMATION

## 2.1. Changes to the Protocol Defined Statistical Analysis Plan

There were no changes or deviations to the originally planned statistical analysis specified in Protocol Amendment 2 (Dated: 18/Jan/2016).

This document contains the RAP amendment 01 which is based on the protocol amendment 2 noted above. RAP amendment 01 revisions primarily include redefining the Screened But Not Enrolled and the Enrolled study populations. These study populations will now be defined as the Screened But Not Evaluable and Evaluable populations. This amendment 01 includes no major changes to the planned analyses. The summary of RAP amendment 01 changes is contained in Appendix 17.

# 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To assess the utility of a BPE/BPO screening tool in conjunction with serum prostate specific antigen (PSA) in finding men confirmed to have BPH on full Urologist assessment of diagnostic test results. | <ul> <li>Proportion of men that are confirmed to have BPH based<br/>on full Urologist assessment of diagnostic test results<br/>among men with a positive result on the BPE/BPO<br/>screening tool (score ≥3) and serum PSA ≥2 ng/mL.</li> </ul> |
| Secondary Objectives | Secondary Endpoints |
| To assess the utility of the BPE/BPO and IPSS screening tools in conjunction with serum PSA in finding men with risk of BPH Progression on full Urologist assessment of diagnostic test results. | <ul> <li>Proportion of men that are confirmed to be a risk for BPH progression based upon full Urologist assessment among men with a positive result on the BPE/BPO, IPSS, BPE/BPO and IPSS, and BPE/BPO or IPSS screening tools and serum PSA ≥2 ng/mL.</li> </ul> |
| To assess the utility of the BPE/BPO and IPSS screening tools in finding men diagnosed with probable BPH¹ as assessed by the GP. | Proportion of men that are diagnosed with probable BPH¹ as assessed by the GP among men with a positive result on the BPE/BPO, IPSS, BPE/BPO and IPSS, and BPE/BPO or IPSS screening tools. |
| To assess the utility of the IPSS screening tool in conjunction with serum PSA in finding men confirmed to have BPH on full Urologist assessment of diagnostic test results. | <ul> <li>Proportion of men that are confirmed to have BPH based<br/>on full Urologist assessment of diagnostic test results<br/>among men with a positive result on the IPSS screening<br/>tool (score ≥8) and serum PSA ≥2 ng/mL.</li> </ul> |
| Compare the utility of the BPE/BPO screening tool with the IPSS screening tool. Probable BPH is the presumptive discression. | Level of agreement (using Kappa statistic for categories) between the BPE/BPO and the IPSS screening tools for selecting men to investigate for BPH. of uriners treat shorts at increase an explorated prostate based on |
| Probable BPH is the presumptive diagnosis | s of urinary tract obstruction from an enlarged prostate based on |

## 2.3. Study Design

## **Overview of Study Design and Key Features**

Description of Visits:

VISIT 1 (primary care clinic)

- Males  $\geq$ 50 years visiting GP for reasons unrelated to the study
- Patient provides informed consent

Eligible to participate

- Inclusion/exclusion criteria confirmation
- Medical history and demography
- BPE/BPO and IPSS screening tools

If subject meets entry criteria, including a positive IPSS (score ≥8) and/or BPE/BPO (score ≥3).

ENROLLED: Subject is enrolled and proceeds to Part I (GP Assessment) of the study. If the GP diagnoses probable BPH, the subject will proceed to Part II (urologist assessment).

PART I: GP Assessment

After being enrolled, complete the following at Visit 1:

- Urinalysis strip test.
  - If strip test is positive, send urine sample to local lab urinalysis.
- PSA blood test
- Additional testing may be performed as per standard of care to assist with a confirmatory diagnosis such as a DRE, however this is not required.

# **Overview of Study Design and Key Features** VISIT 2 (telephone call) GP reviews urinalysis and PSA lab results. Call subject: If lab results show NO probable BPH, then subject will not continue in the study. If PSA lab results show PROBABLE BPH (≥2 ng/mL), subject proceeds to Part II and Visit 3 is scheduled for the urologist assessment. The subjects Does subject have urinary NO participation in the track symptoms? study is concluded YES The subjects Does subject have NO participation in the probable BPH? study is concluded YES Proceed to Part II: Schedule urologist assessment

## **Overview of Study Design and Key Features**

VISIT 3 (Part II – urologist clinic visit)

- Urologist reviews medical history and symptoms
- Brief physical examination
- DRE
- Review previous tests (BPE/BPO screening tool, IPSS screening tool, urinalysis, PSA)



Urologist provides:

- Confirmation of clinical diagnosis of BPH (or confirmation the subject does NOT have BPH).
- Estimate whether the patient is at risk of progression of BPH (PSA≥2.0ng/mL and other tests).
- NOTE: Urologist may need to perform additional diagnostic testing as per standard of care and as needed to assess the BPH diagnosis. This follow-up is not prescribed by this protocol, however, any data collected that is used for the final diagnosis will be entered in the study case report form (CRF). Advice or treatment post study will be discretion of the GP or Urologist.

## **Design Features**

- No investigational study drug is being administered during this study.
- This is a non-randomized, interventional study utilizing a questionnaire-based assessment of men in General Practice. Men who sign the informed consent form and meet the eligibility criteria will be enrolled and complete the Part I diagnostic tests at the GP clinic. If the GP determines that the subject has probable BPH, the subject proceeds to Part II and is scheduled for a Urologist assessment and diagnostic tests to confirm or refute a BPH diagnosis and to assess the risk of progression of BPH.

| Overview of | Overview of Study Design and Key Features |
|---|---|
| Dosing | No investigational study drug is being administered during this study. |
| Treatment<br>Assignmen<br>t | <ul> <li>Subjects are not randomized or dispensed study treatment.</li> <li>Approximately 1,500 males presenting to a GP with a primary complaint other than LUTS will be screened for probable BPH to yield 500 subjects being referred to a Urologist.</li> </ul> |
| Interim<br>Analysis | No interim analyses are planned for this study. |

## 2.4. Statistical Hypotheses

The primary endpoint is defined as the proportion of men confirmed to have BPH based on full Urologist diagnostic testing in men with a positive result on the BPE/BPO screening tool and a probable BPH assessment by GP. Primary endpoint summaries will be descriptively presented in terms of the calculated proportion, described below, and a 95% confidence interval on the proportion. Formal hypothesis testing will not be conducted in terms of the primary and secondary endpoint proportions.

#### 3. PLANNED ANALYSES

## 3.1. Interim Analyses

No interim analyses are planned for this study.

# 3.2. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All subjects have either completed, or withdrawn from, the study, as defined in the protocol.
- 2. All required database cleaning activities have been completed and final database release and database freeze has been declared by Data Management.

The primary database freeze, using standard Data Management practices, will occur after the last subject completes Visit 3. Statistical analysis and reporting will be in terms of this primary database freeze and will be referred to as the 'Final Analysis' or primary 'Statistical Analysis Complete' (SAC).

## 4. ANALYSIS POPULATIONS

No investigational study drug is being administered during this study.

This is a non-randomized, interventional study utilizing a questionnaire-based assessment of men in general practice, therefore the populations are not defined in the traditional sense. The following populations will be used on this study.

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Screened | Comprised of all subjects who are screened for eligibility. | <ul> <li>Study Population</li> <li>Efficacy (agreement<br/>between BPE/BPO<br/>and IPSS)</li> </ul> |
| Screened But Not Evaluable | Comprised of all subjects who are screened for<br>eligibility, but do not qualify for the Evaluable<br>Population. | <ul><li>Study Population</li><li>Safety (Adverse<br/>Events Listing)</li></ul> |
| Evaluable | <ul> <li>Comprised of all subjects who meet the entry<br/>criteria, including a positive IPSS screening<br/>result (score ≥8) and/or a positive BPE/BPO<br/>screening result (score ≥3).</li> </ul> | <ul><li>Study Population</li><li>Efficacy</li><li>Safety</li></ul> |

**NOTES:** Please refer to Appendix 15: List of Data Displays which details the population to be used for each display being generated.

#### 4.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarized and listed.

#### 4.1.1. Inclusion / Exclusion Criteria Deviations

All inclusion / exclusion criteria deviations which are recorded on the inclusion / exclusion screens of the eCRF will be summarized. The tabular summaries will be in terms of number and percent of Screened But Not Evaluable Subjects violating any criterion and violating each criterion.

Listings of inclusion / exclusion criteria deviations will be produced for Screened But Not Evaluable subjects.

#### 4.1.2. Important Protocol Deviations

Protocol deviations identified during the study will be tracked and reviewed by the study team in accordance with SOP-130050 and the FDC116114 Protocol Deviation Management Plan (PDMP). Prior to the final database lock and data analysis for the clinical study report (CSR), the FDC116114 Study team will determine whether any subjects will be excluded from the summary of important protocol deviations as specified in the reporting and analysis plan. Protocol deviation data entered into the eCRF (InForm) will be extracted and processed as a SAS dataset with identifiers for important protocol deviations. Subjects with important protocol deviations will be summarized and

discussed, and the CSR listings will include a list of important protocol deviations occurring in the study; listings of all protocol deviations will be available for regulators if requested.

- Data will be reviewed prior to freezing the database to ensure all important deviations are captured and categorized on the protocol deviations dataset.
- This dataset will be the basis for the summaries and listings of protocol deviations.

Important Deviations will be summarized and listed for Evaluable subjects. The tabular summary will be in terms of number and percent of subjects with any Important Deviations and with each Important Deviation. Summaries will be output by the eCRF categories for the Evaluable subjects and by the following screening tool categories: IPSS≥8, BPE/BPO≥3, IPSS≥8 and BPE/BPO≥3, and IPSS≥8 or BPE/BPO≥3. The eCRF categories are standardized for this study; examples are provided in the tabular summary shells.

Listings of important protocol deviations will be produced for Evaluable subjects.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

Table 1 provides an overview of appendices within the RAP for outlining general considerations for data analyses and data handling conventions. A full set of appendices is provided in Section 11.

Table 1 Overview of Appendices

| Section | Component |
|---|---|
| 11.1 | Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population |
| 11.2 | Appendix 2: Time & Events |
| 11.3 | Appendix 3: Assessment Windows |
| 11.4 | Appendix 4: Treatment States and Phases |
| 11.5 | Appendix 5: Data Display Standards & Handling Conventions |
| 11.6 | Appendix 6: Derived and Transformed Data |
| 11.7 | Appendix 7: Premature Withdrawals & Handling of Missing Data |
| 11.8 | Appendix 8: Adverse Event Time Periods and Special Adverse Event Definitions |
| 11.9 | Appendix 9: Values of Potential Clinical Importance |
| 11.10 | Appendix 10: Multicenter Studies |
| 11.11 | Appendix 11: Examination of Covariates, Subgroups & Other Strata |
| 11.12 | Appendix 12: Multiple Comparisons & Multiplicity |
| 11.13 | Appendix 13: Model Checking and Diagnostics for Statistical Analyses. |
| 11.14 | Appendix 14: Abbreviations and Trademarks |
| 11.15 | Appendix 15: List of Data Displays |
| 11.16 | Appendix 16: Example Mock Shells for Data Displays |
| 11.17 | Appendix 17: Amendment 01 Revisions |

## 6. STUDY POPULATION ANALYSES

## 6.1. Overview of Planned Analyses

The study population analyses will be based on the Evaluable subjects, unless otherwise specified.

Table 2 provides an overview of the planned study population summaries and listings, with full details of planned data displays being presented in Appendix 15: List of Data Displays. All summaries will be presented by the following categories: IPSS≥8, BPE/BPO≥3, IPSS≥8 and BPE/BPO≥3, and IPSS≥8 or BPE/BPO≥3, unless otherwise noted.

Formal hypothesis testing will not be performed in terms of the study population data.

Table 2 Overview of Planned Study Population Analyses

| Display Type | Data Displays Generated | | |
|---|---|---|---|
| | Table | Figure | Listing |
| Subject Accountability | | | |
| Numbers of Subjects, including Screened, Screened But | Υ | | |
| Not Evaluable, and Evaluable | I | | |
| Number of Subjects, including: Evaluable, Evaluable with | | | |
| PSA Values (<2 or ≥2), GP Assessments, and Urologist | Y | | Υ |
| Assessments | | | |
| Subject Disposition | | | |
| Overall Disposition | Y | | Υ |
| Subject Withdrawals | Υ | | Υ |
| Discontinuation by Visit | Υ | | |
| Inclusion / Exclusion Criteria Deviations (Screened But Not | Y | | Y |
| Evaluable Subjects) | • | | ı |
| Important Protocol Deviations | Υ | | Υ |
| Demographic Characteristics | | | |
| Demographic Characteristics | Υ | | Υ |
| Race | Υ | | Υ |
| Medical Conditions and Concomitant Medications | | | |
| Medical Conditions by Body System | Υ | | Υ |
| Surgical / Diagnostic Procedures | Υ | | Υ |
| Concomitant Medications | Υ | | Υ |
| Diagnostic Tests and Questionnaires | | | |
| PSA | Y | | |
| IPSS and BPE/BPO | Y | | |

#### NOTES:

- Y = Yes display generated.
- There are no planned Study Population Figures.

## 6.2. Subject Accountability

Summaries for the following will be produced in terms of total number overall:

- All Screened Subjects
- All Evaluable Subjects

Evaluable subjects include those subjects who met all inclusion and exclusion criteria including a positive IPSS (score≥8) and/or BPE/BPO (score≥3). Summaries for the Screened and Evaluable subjects will also be presented by country, and separately by country and center.

A summary table will be produced for the screened subjects and will contain the following:

- Number of subjects who were sScreened but not Evaluable
- Number of subjects who were Evaluable

A summary of screened subjects by country, and separately by country and center will also be presented.

A summary table will be produced for the Evaluable subjects and will contain the following:

- All Evaluable Subjects (IPSS\ge 8 or BPE/BPO\ge 3)
- Evaluable Subjects with PSA<2.0ng/mL
- Evaluable Subjects with PSA\ge 2.0ng/mL
- Evaluable Subjects with Any GP Assessment of BPH
- Evaluable Subjects with GP Assessment of BPH="Yes"
- Evaluable Subjects with GP Assessment of BPH="No"
- Evaluable Subjects with GP Assessment of BPH="Yes" and Urologist Assessment of BPH
- Evaluable Subjects with GP Assessment of BPH="Yes" and Urologist Assessment of BPH="Yes"
- Evaluable Subjects with GP Assessment of BPH="Yes" and Urologist Assessment of BPH="No"
- Evaluable Subjects with GP Assessment of BPH="Yes" and Any Urologist Risk Assessment of BPH Progression
- Evaluable Subjects with GP Assessment of BPH="Yes" and Urologist Risk Assessment of BPH Progression="Yes"
- Evaluable Subjects with GP Assessment of BPH="Yes" and Urologist Risk Assessment of BPH Progression="No"

An overall summary and the data above will also be presented by country, and separately by country and center for the Evaluable subjects.

## 6.3. Subject Disposition

A subject may withdraw from the study at any time at the investigator's discretion or at the request of the subject.

The reason for study withdrawal is recorded in the eCRF for Evaluable subjects who prematurely withdrew from the study prior to completing Visits 1, 2, and 3. A tabular summary will be produced for number and percentage of subjects prematurely withdrawing from the study, overall and by reason. Additional tabular summaries will be produced by Visit (overall and by reason) for subjects withdrawing from the study. For these summaries, the percentages are calculated using the number of subjects in each of the categories (IPSS≥8, BPE/BPO≥3, IPSS≥8 and BPE/BPO≥3, and IPSS≥8 or BPE/BPO≥3) as the denominators.

Listings will be produced for subject disposition and reason for withdrawal and will include key accountability data including study status, completion or withdrawal date, all visit dates, and the primary reason for premature withdrawal.

## 6.4. Demographic Characteristics

The following demographic characteristics will be summarized for the Screened But Not Evaluable and Evaluable subjects; summaries for the Evaluable subjects will be repeated by country, and separately by country and center:

- Sex
- Age in years
- Age categories (years):  $<65, \ge 65, <75, \ge 75$
- Race (Evaluable subjects only)

Listings will be produced for sex, age, and race (Evaluable subjects only). Race information will not be presented in tables or listings for subjects who were enrolled in the study in France.

# 6.5. Medical Conditions, Surgical Procedures, and Concomitant Medications

The following medical conditions and surgical procedures are GSK standardized data collections and/or are of interest in terms of the Evaluable subjects, and will be summarized in tabular and listing formats. The number and percentage of subjects reporting having each medical condition or surgical procedure will be included in the summary. Tabular summaries of surgical procedures will be presented for screening and post-screening visits.

#### **Medical Conditions**

- Cardiovascular Risk Factors
  - o Angina Pectoris
  - Myocardial Infarction

- Stroke
- Diabetes
- Hypertension
- o Hyperlipidemia
- Urinary Conditions
  - o Incomplete Urination
  - Unable to Urinate
  - Urination Difficulty
  - Micturition Disorder
  - o Increased Urinary Frequency
  - o Recurrent Urinary Tract Infection
  - Hematuria
  - o Urinary Incontinence Surgery
  - Urethral Stricture
  - Urine Flow Decreased
  - o Post Void Dribbling
  - o Nocturia
  - Urinary Calculus
  - o Bladder Neoplasm/Tumor

#### **Surgical Procedures**

- Cystoscopy
- Transrectal Ultrasound
- Prostate Biopsy
- Ultrasound Abdomen
- Computerized Tomogram Abdomen
- Computerized Tomogram Pelvis
- Nuclear MRI Abdominal
- Pelvic MRI
- Renal Scan
- Bladder Scan
- Abdominal X-Ray
- Other

Concomitant medication data are collected on eCRF log forms and will be coded using the GSKDrug dictionary. Concomitant medications will be defined as any medication documented as such in the database, irrespective of start or stop dates or ongoing status.

A summary of concomitant medications will be provided. The number and percentage of subjects reporting the use of each concomitant medication will be summarized and will include ATC Level I and ingredient. A listing of the collected concomitant medications by country and center will be provided. A listing of the relationship between the ATC Level I, ingredient, and verbatim text for concomitant medications will also be provided.

## 6.6. Diagnostic Tests and Questionnaires

The IPSS screening tool is completed at the screening visit. The total IPSS score is the sum of the 7 individual questions. The total IPSS score will be summarized by N, Mean, Standard Deviation, Median, Minimum, and Maximum. The number and percentage of subjects with total IPSS scores will also be summarized categorically using the following categories:  $\langle 8, 8-19, \rangle 19$ .

The BPE/BPO screening tool is completed at the screening visit. The total BPE/BPO score is the sum of the 3 individual questions. The total BPE/BPO score will be summarized by N, Mean, Standard Deviation, Median, Minimum, and Maximum. The number and percentage of subjects with total BPE/BPO scores will also be summarized categorically using the following categories: <3, 3-6, >6.

Serum PSA samples are scheduled at the screening visit after the subject is enrolled. Serum PSA will be summarized by N, Mean, Standard Deviation, Median, Minimum, and Maximum. The number and percentage of subjects with serum PSA data will also be summarized categorically using the following categories: <2, 2-9, >9.

The IPSS, BPE/BPO, and PSA data described above will also be summarized by country, and separately by country and center.

## 7. PRIMARY STATISTICAL ANALYSES

## 7.1. Primary Efficacy Analyses

## 7.1.1. Overview of Planned Primary Efficacy Analyses

The primary endpoint is defined as the proportion of men confirmed to have BPH based on full Urologist diagnostic testing among men with a positive result on the BPE/BPO screening tool (score  $\geq$ 3) and serum PSA  $\geq$ 2 ng/mL. The BPE/BPO questionnaire consists of three questions each with a score ranging from 0 to 5. This questionnaire is administered at the screening visit (Visit 1).

BPE/BPO (also called the BPE/BPO total score) is the sum of the three questions. BPE/BPO summaries will be in terms of the total (score); exceptions will be noted such as for supporting summaries of individual questions. For calculation of the BPE/BPO total, missing individual responses will not be imputed.

The primary efficacy analyses will be based on the Evaluable subjects, unless otherwise specified. Table 3 provides an overview of the planned BPE/BPO summaries and primary efficacy analyses, with full details of data displays being presented in Appendix 15: List of Data Displays.

Table 3 Overview of Planned Primary Efficacy Analyses

| | | | | | Abso | olute | |
|---|---|---|---|---|---|---|---|
| Endpoint | Stats Analysis | | Summary | | Individual | | |
| Liidpoliit | T | F | L | T | F | F | L |
| Proportion of Men with | <b>BPH Based</b> | on full Uro | logist Diag | nosis and I | BPE/BPO So | core (≥3) | |
| Primary Analysis | <b>Y</b> [1] | | | | | | |
| Supporting Data for Pri | mary Endp | oint | | | | | |
| BPE/BPO Individual | | | | | | | |
| and Total Scores at | | | | <b>Y</b> [2] | | | <b>Y</b> [2] |
| Visit 1 | | | | | | | |
| Summary of PSA | | | | | | | |
| Values | | | | <b>Y</b> [3] | | | <b>Y</b> [3] |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
  - 1. Primary efficacy analyses are presented within this table; details of the analysis are in the following section.
  - 2. Individual BPE/BPO question 1-3 responses and total scores support the primary analysis; total scores are also presented by country, and separately by country and center.
  - 3. The PSA summary data supports the primary analysis; the PSA data Tables and Listings appear with the Safety Tables and Listings.

## 7.1.2. Planned Primary Efficacy Statistical Analyses

## **Primary Statistical Analyses**

## Endpoint(s)

- Proportion of men that are confirmed to have BPH based on full Urologist assessment of diagnostic test results among men with a positive result on the BPE/BPO screening tool (score ≥3) and serum PSA ≥2 ng/mL.
- Primary endpoint summaries will be descriptively presented in terms of the calculated proportion, described below, and 95% confidence interval on the proportion. Formal hypothesis testing will not be conducted.

| Tool | Proportion | Numerator | Denominator |
|---|---|---|---|
| BPE/BPO | BPH diagnosis by Urologist based upon BPE/BPO screening tool (score≥3) and serum PSA ≥2 ng/mL. | Number of subjects<br>diagnosed with BPH<br>based upon a BPH<br>assessment by<br>Urologist. | Number of subjects with a positive result on the BPE/BPO screening tool (score≥3) and serum PSA ≥2 ng/mL and a BPH assessment by Urologist. |

Table 3 provides an overview of the planned summaries and primary efficacy analyses. A list
of planned data displays is in Appendix 15: List of Data Displays.

## **Model Specification**

 No models were used during the statistical analysis; proportions and confidence intervals were computed.

## **Model Checking & Diagnostics**

Not Applicable

## **Model Results Presentation**

Not Applicable

#### Sensitivity and Supportive Statistical Analyses

Not Applicable

## 8. SECONDARY STATISTICAL ANALYSES

# 8.1. Secondary Efficacy Analyses

# 8.1.1. Overview of Planned Secondary Efficacy Analyses

The secondary efficacy analyses will be based on the Evaluable subjects, unless otherwise specified. Table 4 provides an overview of the planned secondary efficacy analyses, with further details of data displays being presented in Appendix 15: List of Data Displays.

Table 4 Overview of Planned Secondary Efficacy Analyses

| | | | | Absolute | | | |
|---|---|---|---|---|---|---|---|
| | ; | Stats Analys | is | Sun | nmary | | ridual |
| Endpoint | T | F | L | Т | F | F | L |
| IPSS | | | | | | | |
| Total and individual | | | | Υ | | | Υ |
| scores at Visit 1 | | | | | | | |
| <b>BPH-Related Health Sta</b> | atus | | | | | | |
| Scores at Visit 1 | | | | Υ | | | Υ |
| BPE/BPO | | | • | | | | • |
| Total and individual | | | | Υ | | | Υ |
| scores at Visit 1 | | | | | | | |
| Summary of BPH Diagr | nosis by U | rologist <sup>[1]</sup> , S | ummary of | <b>BPH Progr</b> | ession Risk | by Urologis | t, and |
| Summary of Probable I | | | , | J | | , , | |
| Based upon BPE/BPO | | | | | | | |
| score (≥3) | Υ | | | | | | |
| Based upon IPSS | | | | | | | |
| score (≥8) | Υ | | | | | | |
| Based upon IPSS | | | | | | | |
| score (≥8) or | Υ | | | | | | |
| BPE/BPO score (≥3) | | | | | | | |
| Based upon IPSS | | | | | | | |
| score (≥8) and | Υ | | | | | | |
| BPE/BPO score (≥3) | | | | | | | |
| Summary of Subjects | Who Disco | ntinued Fro | m the Stud | v Before th | e GP Was A | ble to Asses | s the |
| Presence of Probable E | | | | | | | |
| <b>Urologist Visit, Among</b> | Subjects V | Who Were E | ligible for S | Such a Visit | | | |
| Based upon BPE/BPO | | | | | | | |
| score (≥3) | Υ | | | | | | |
| Based upon IPSS | | | | | | | |
| score (≥8) | Υ | | | | | | |
| Based upon IPSS | | | | | | | |
| score (≥8) or | Υ | | | | | | |
| BPE/BPO score (≥3) | | | | | | | |
| Based upon IPSS | | | | | | | |
| score (≥8) and | Υ | | | | | | |
| BPE/BPO score (≥3) | | | | | | | |

| | | | | | Abso | olute | |
|---|---|---|---|---|---|---|---|
| | S | tats Analysis | 3 | Summary | | Individual | |
| Endpoint | T | F | L | T | F | F | L |
| BPE/BPO and IPSS | BPE/BPO and IPSS | | | | | | |
| Summary of | | | | | | | |
| agreement between | Υ | | | | | | |
| screening tools (Kappa | | | | | | | |
| statistic) | | | | | | | |
| Figures (All Evaluable S | Subjects) | | | | | | |
| Plot of IPSS Scores | | | | | | | |
| versus BPE/BPO | | | | | Υ | | |
| Scores at Visit 1 | | | | | | | |
| Plot of IPSS Scores | | | | | | | |
| versus PSA Values at | | | | | Υ | | |
| Visit 1 | | | | | | | |
| Plot of BPE/BPO | | | | | | | |
| Scores versus PSA | | | | | Υ | | |
| Values at Visit 1 | | | | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
  - 1. Summary of BPH diagnosis by the Urologist based upon the BPE/BPO screening tool (score ≥3) is a Primary Endpoint and is not included in the Secondary Endpoint analysis.

# 8.1.2. Planned Secondary Efficacy Statistical Analyses

# **Primary Statistical Analyses**

#### Endpoint(s)

Secondary endpoints and other measures of interest are defined in terms of proportions for each: probable BPH diagnosis by GP, BPH diagnosis by Urologist, and BPH progression risk by Urologist along with use of 1) BPE/BPO screening tool and 2) IPSS screening tool. The 95% confidence intervals (calculated using the exact (Clopper-Pearson) method) for these proportions will be presented.

| Tool | Proportion | Numerator | Denominator |
|---|---|---|---|
| BPE/<br>BPO | BPH Progression Risk by<br>Urologist based upon<br>BPE/BPO screening tool<br>(score ≥3) and serum<br>PSA ≥2 ng/mL | Number of subjects<br>diagnosed with BPH<br>progression risk by<br>Urologist | Number of subjects with a positive result on the BPE/BPO screening tool (score ≥3) and serum PSA ≥2 ng/mL and a BPH progression risk assessment by Urologist |
| BPE/<br>BPO | Probable BPH Diagnosis<br>by GP based upon<br>BPE/BPO screening tool<br>(score ≥3) | Number of subjects<br>diagnosed with 'probable<br>BPH' by GP | Number of subjects with a positive result on the BPE/BPO screening tool (score ≥3) and a BPH assessment by GP |

#### **Primary Statistical Analyses**

| Secor | Secondary Endpoints: Proportions only in terms of the IPSS screening tool | | |
|---|---|---|---|
| Tool | Proportion | Numerator | Denominator |
| IPSS | BPH Diagnosis by<br>Urologist based upon<br>IPSS (score ≥8) and<br>serum PSA ≥2 ng/mL | Number of subjects diagnosed with BPH based upon BPH assessment by Urologist. | Number of subjects with a positive result on the IPSS (score ≥8) and serum PSA ≥2 ng/mL and a BPH assessment by Urologist |
| IPSS | BPH Progression Risk by<br>Urologist based upon<br>IPSS (score ≥8) and<br>serum PSA ≥2 ng/mL | Number of subjects<br>diagnosed with BPH<br>progression risk by<br>Urologist | Number of subjects with a positive result on the IPSS (score ≥8) and serum PSA ≥2 ng/mL and a BPH progression risk assessment by Urologist |
| IPSS | Probable BPH Diagnosis<br>by GP based upon IPSS<br>(score ≥8) | Number of subjects<br>diagnosed with 'probable<br>BPH' by GP | Number of subjects with a positive result on the IPSS (score ≥8) and a BPH assessment by GP |

- Additional summaries, proportions and related 95% confidence intervals, will be generated as
  outlined above, but in terms of a positive result for both the BPE/BPO and the IPSS screening
  tools and separately for either the BPE/BPO or IPSS screening tools.
- Another secondary endpoint of this study is to assess the level of agreement (via the kappa statistic) between the BPE/BPO and/or IPSS screening tools for selecting men to investigate for BPH. The number and proportion of subjects with a positive or with a negative response to both the BPE/BPO and IPSS screening tools at screening will be summarized.
- The kappa coefficient will be characterized as proposed by Landis and Koch (Landis, 1977) with <0 indicating no agreement, 0-0.20 as slight, 0.21-0.40 as fair, 0.41-0.60 as moderate, 0.61-0.80 as substantial, and 0.81 1 as almost perfect agreement.</li>
- The proportion of subjects who discontinued from the study before the GP was able to assess
  the presence of probable BPH will be summarized. The proportion of subjects who withdrew
  from the study before a Urologist visit, among subjects with a probable GP BPH diagnosis will
  be summarized.

#### **Model Specification**

 No models were used during the statistical analysis; proportions and confidence intervals were computed.

## **Model Checking & Diagnostics**

Not Applicable

#### **Model Results Presentation**

Not Applicable

## Sensitivity and Supportive Statistical Analyses

Not Applicable

#### 8.1.2.1. IPSS Screening Tool

The IPSS screening tool is completed at the screening visit (Visit 1). The total IPSS score is the sum of the 7 individual questions. The total IPSS score will be summarized by N, Mean, Standard Deviation, Median, Minimum, and Maximum for each of the following:

- All Evaluable Subjects (IPSS\ge 8 or BPE/BPO\ge 3)
- Evaluable Subjects with PSA<2.0ng/mL
- Evaluable Subjects with PSA≥2.0ng/mL
- Evaluable Subjects with Any GP Assessment of BPH
- Evaluable Subjects with GP Assessment of BPH="Yes"
- Evaluable Subjects with GP Assessment of BPH="No"
- Evaluable Subjects with GP Assessment of BPH="Yes" and Urologist Assessment of BPH
- Evaluable Subjects with GP Assessment of BPH="Yes" and Urologist Assessment of BPH="Yes"
- Evaluable Subjects with GP Assessment of BPH="Yes" and Urologist Assessment of BPH="No"
- Evaluable Subjects with GP Assessment of BPH="Yes" and Any Urologist Risk Assessment of BPH Progression
- Evaluable Subjects with GP Assessment of BPH="Yes" and Urologist Risk Assessment of BPH Progression="Yes"
- Evaluable Subjects with GP Assessment of BPH="Yes" and Urologist Risk Assessment of BPH Progression="No"

The total IPSS score will be presented by the following categories: IPSS\ge 8, BPE/BPO\ge 3, IPSS\ge 8 and BPE/BPO\ge 3, and IPSS\ge 8 or BPE/BPO\ge 3. The total IPSS score data will also be presented by country, and separately by country and center.

A listing of the IPSS individual and total scores will be presented.

#### 8.1.2.2. BPH-Related Health Status

BPH-Related Health Status (BHS) is collected as Question 8 on the IPSS questionnaire and ranges from 0 to 6. The IPSS questionnaire is administered, and thus BHS is collected, at the screening visit (Visit 1). The total number, as well as the number and percentage of subjects experiencing quality of life symptoms, will be provided.

BPH-Related Health Status values will be presented by the following categories: IPSS\geq 8, BPE/BPO\geq 3, IPSS\geq 8 and BPE/BPO\geq 3, and IPSS\geq 8 or BPE/BPO\geq 3. The BPH-Related Health Status data will also be presented by country, and separately by country and center.

A listing of the BPH-Related Health Status individual scores will be presented.

#### 8.1.2.3. BPE/BPO Screening Tool

The BPE/BPO screening tool is completed at the screening visit (Visit 1). The total BPE/BPO score is the sum of the 3 individual questions. The total BPE/BPO score will be summarized by N, Mean, Standard Deviation, Median, Minimum, and Maximum for each of the following:

- All Evaluable Subjects (IPSS\ge 8 or BPE/BPO\ge 3)
- Evaluable Subjects with PSA<2.0ng/mL
- Evaluable Subjects with PSA≥2.0ng/mL
- Evaluable Subjects with Any GP Assessment of BPH
- Evaluable Subjects with GP Assessment of BPH="Yes"
- Evaluable Subjects with GP Assessment of BPH="No"
- Evaluable Subjects with GP Assessment of BPH="Yes" and Urologist Assessment of BPH
- Evaluable Subjects with GP Assessment of BPH="Yes" and Urologist Assessment of BPH="Yes"
- Evaluable Subjects with GP Assessment of BPH="Yes" and Urologist Assessment of BPH="No"
- Evaluable Subjects with GP Assessment of BPH="Yes" and Any Urologist Risk Assessment of BPH Progression
- Evaluable Subjects with GP Assessment of BPH="Yes" and Urologist Risk Assessment of BPH Progression="Yes"
- Evaluable Subjects with GP Assessment of BPH="Yes" and Urologist Risk Assessment of BPH Progression="No"

The total BPE/BPO score will be presented by the following categories: IPSS≥8, BPE/BPO≥3, IPSS≥8 and BPE/BPO≥3, and IPSS≥8 or BPE/BPO≥3. The total BPE/BPO score data will also be presented by country, and separately by country and center.

A listing of the BPE/BPO individual and total scores will be presented.

## 8.2. Safety Analyses

## 8.2.1. Overview of Planned Analyses

Safety summaries and analyses are reported in terms of the following data classifications: adverse events, clinical laboratory assessments (urinalysis), total serum prostate specific antigen (PSA), and digital rectal examination (DRE).

All safety analyses will be performed using the Evaluable subjects unless otherwise specified in text or data display shells. Applicable safety analysis and reporting definitions and presentations within "Program Safety Analysis Plan (PSAP, 2016) for GI198745 (dutasteride) and GSK2285985 (fixed dose combination of dutasteride [GI198745] and tamsulosin [GI138525]" are utilized within this RAP, with any deviations noted.

Table 5 provides an overview of the planned adverse event tabular summaries. A list of planned data displays is in Appendix 15: List of Data Displays.

Reference Section 4 (Analysis Populations) and Appendix 6 (Derived and Transformed Data) for supporting definitions on all below subsections.

Table 5 Overview of Planned Safety Analyses

| Adverse Event Types, High Level | | | | | |
|---|---|---|---|---|---|
| - | | | | Leading to W/D | |
| | Any | Non-Serious | Serious | from Study | Fatal |
| By Type | | 3.1 (5 above | categories, excluding | g Non-Serious) | |
| | | | 3.11 | 3.17 | 3.16 |
| Overall | 3.2 | 3.3 | 3.14 | 3.18 | |
| By Age (<65, ≥65, <75, | 3.4 | | 3.12 | | |
| ≥75) | 3.5 | | 3.13 | | |
| By Country; By | 3.6 | | 3.14 | | |
| Country and Center | 3.7 | | 3.15 | | |
| By Maximum Intensity | 3.8 | | | | |
| Most Common | 3.9 | 3.10 | | | |
| Sexual and Breast Adve | erse Events of Spec | ial Interest | | | |
| MedDRA | | | 3.19 | | |
| <b>Prostate Cancer Advers</b> | se Event of Special | Interest | | | |
| Prostate Cancer | | | 3.20 | | |
| Overall | | | | | |
| Cardiovascular Adverse | Cardiovascular Adverse Events of Special Interest | | | | |
| MedDRA | 3.21 | | | | |
| Infrequent Tier 1 Advers | Infrequent Tier 1 Adverse Events of Special Interest | | | | |
| MedDRA | | | 3.22 | | |

#### NOTES:

• Summaries are in terms of 'starting on or after enrollment' (defined in Appendix 6) unless otherwise noted.

#### 8.2.2. Adverse Events

Adverse events (AEs) will be coded using the MedDRA (Medical Dictionary for Regulatory Activities) coding dictionary. As specified in the protocol, disease related events will not be reported as AEs or serious adverse events (SAEs) unless the investigator assesses the event as more severe than expected for the subject's condition. A mapping of the MedDRA primary system organ class and preferred term to which each verbatim term has been coded will be provided in a listing.

Adverse events (AEs) are to be recorded on the electronic case report form (eCRF) from the time of enrollment until the end of the study period (completion of Visits 1, 2, and 3). Serious AEs (SAEs) are to be recorded from the time of informed consent. Any SAEs assessed as related to study participation or related to a GSK concomitant medication, will be recorded from the time a subject consents to participate in the study up to the completion of the subject's final visit. The investigator will monitor all AEs/SAEs that are ongoing until resolution or stabilization of the event, or until the subject is lost to follow-up. Adverse events summaries will include non-serious as well as serious AEs.

The number of post-enrollment adverse events, the number and the percentage of subjects reporting any post-enrollment AE will be summarized for the following:

- All AEs
- Serious AEs
- AEs leading to withdrawal from study
- Fatal AEs

Total number of adverse events reported in the study as well as the number and percentage of subjects reporting at least one AE will be provided. Total number of AEs as well as the number and percentage of subjects reporting each AE will be reported by primary system organ class and preferred term. Non-serious post-enrollment AEs will be summarized. A summary of post-enrollment AEs will be provided by age group (<65, ≥65, <75, ≥75 years), by country, and separately by country and center.

A summary of post-enrollment AEs will also be provided by maximum intensity. If the same AE occurs on multiple occasions in the same subject, the AE with the highest intensity will be presented. Intensity will be categorized as mild, moderate, or severe; a category for missing/not applicable intensity will be included.

The most common AEs (Tier 2 events) are defined as those preferred terms occurring in at least 5% of the subjects (non-rounded). The total number of events as well as the number and percentage of subjects reporting at least one most common AE preferred term starting post-enrollment will be provided. The total number of events as well as the number and percentage of subjects reporting at least one non-serious most common AE preferred term starting post-enrollment will also be provided. Individual subject listings of all adverse events for the Screened But Not Evaluable and for the Evaluable subjects will be presented.

#### 8.2.3. Deaths and Serious Adverse Events

Total number of serious adverse events as well as the number and percentage of subjects reporting at least one serious AE will be provided. Total number of serious adverse events as well as the number and percentage of subjects reporting each serious AE will be reported by primary system organ class and preferred term. A summary of postenrollment serious AEs will be provided by age group ( $<65, \ge65, <75, \ge75$ ), by country, and separately by country and center. A summary of all post-enrollment fatal AEs will be provided.

Individual subject listings of all non-fatal serious AEs and a separate listing of all fatal AEs will be provided. The listing will indicate the timing of the serious AE with respect to enrollment date.

# 8.2.4. Adverse Events Leading to Withdrawal From the Study and Other Significant Adverse Events

## 8.2.4.1. Adverse Events Leading to Withdrawal from the Study

A summary of adverse events starting post-enrollment and leading to withdrawal from the study will be provided for the following categories:

- All AEs
- Serious AEs

Subject listings of AEs leading to withdrawal from the study will be provided. The listings will indicate the timing of the AE with respect to enrollment start date.

#### 8.2.4.2. Adverse Events of Special Interest

Tier 1 adverse events of special interest are pre-specified adverse event preferred terms for which there are predefined hypotheses about the existence of a potential occurrence. These events include the following:

- Sexual and breast events
- Prostate cancer
- Cardiovascular events
- Infrequent events

Summaries for these events are specified in the following sections and will be based on post-enrollment AEs unless otherwise indicated. A mapping of the MedDRA primary system organ class and preferred term to which each verbatim term in the special interest AE categories has been coded will be provided in a listing.

#### 8.2.4.3. Sexual and Breast Tier 1 Adverse Events of Special Interest

Altered (decreased) libido, impotence, ejaculation disorders, and breast disorders, will be defined as sexual and breast adverse events of special interest. Two subgroups of breast disorders (breast disorders: breast enlargement, and breast disorders: breast tenderness) are of special interest. MedDRA system organ class and preferred terms included in these special interest adverse events are defined in Appendix 8, Table A.

Total number of, as well as number and percentage of the subjects experiencing, sexual and breast adverse events of special interest will be provided.

Listings of sexual and breast adverse events of special interest will be provided.

#### 8.2.4.4. Prostate Cancer Adverse Events of Special Interest

Prostate cancer will be defined as an adverse event of special interest. MedDRA preferred terms and codes included in this special interest adverse event are defined in Appendix 8, Table B. Prostate cancer events will be summarized separately following the same format done for sexual and breast special interest AEs described above.

Listings of prostate cancer adverse events of special interest will be provided.

#### 8.2.4.5. Cardiovascular Adverse Events of Special Interest

Cardiovascular adverse events of special interest will be defined as those included in the following six categories: acute coronary syndrome, ischemic coronary artery disorders/atherosclerosis, ischemic cerebrovascular events, cardiac failure, cardiac arrhythmias, and peripheral vascular disease. MedDRA preferred terms and codes included in these special interest adverse events are defined in Appendix 8, Table C. Total number of cardiovascular events as well as the number and percentage of subjects experiencing cardiovascular events will be provided.

Listings of cardiovascular adverse events of special interest will be provided.

#### 8.2.4.6. Infrequent Tier 1 Adverse Events of Special Interest

Infrequent Tier 1 adverse events of special interest will be defined as those included in the following categories:

- Breast cancer
- Potential for decreased male fertility due to effects on sperm/semen characteristics
- Interference with formation of external genitalia in a male fetus if a woman carrying a male fetus is exposed to dutasteride
- Hair changes
- Allergic reactions
- Depressed mood
- Testicular pain and swelling
- Intraoperative floppy iris syndrome
- Orthostasis
- Priapism
- Stevens-Johnson syndrome
- Atrial fibrillation, tachycardia, arrhythmias

MedDRA preferred terms and codes included in these special interest adverse events are defined in Appendix 8, Table D. Total number of infrequent Tier 1 events as well as the number and percentage of subjects with infrequent Tier 1 events will be provided.

Listings of infrequent Tier 1 adverse events of special interest will be provided.

## 8.2.5. Clinical Laboratory Assessments

A urine strip test (dipstick) will be performed at screening for all Evaluable subjects (Visit 1). If the dipstick is positive, the urine sample will be submitted to the local laboratory for urinalysis. The urine microscopy values assessed on the urine sample will include the following parameters:

- Urine Protein
- Urine Glucose
- Urine RBC
- Urine WBC

The overall number of subjects tested and the number and percentage of subjects with positive /negative results will be presented by the following categories: IPSS≥8, BPE/BPO≥3, IPSS≥8 and BPE/BPO≥3, and IPSS≥8 or BPE/BPO≥3. The urinalysis data will also be presented by country, and separately by country and center.

A listing of the urinalysis data will be provided.

#### 8.2.6. Serum PSA

Serum PSA samples are scheduled at the screening visit (Visit 1) after the subject is enrolled. Serum PSA will be summarized by N, Mean, Standard Deviation, Median, Minimum, and Maximum for each of the following:

- All Evaluable Subjects (IPSS\ge 8 or BPE/BPO\ge 3)
- Evaluable Subjects with PSA<2.0ng/mL
- Evaluable Subjects with PSA\ge 2.0ng/mL
- Evaluable Subjects with Any GP Assessment of BPH
- Evaluable Subjects with GP Assessment of BPH="Yes"
- Evaluable Subjects with GP Assessment of BPH="No"
- Evaluable Subjects with GP Assessment of BPH="Yes" and Urologist Assessment of BPH
- Evaluable Subjects with GP Assessment of BPH="Yes" and Urologist Assessment of BPH="Yes"
- Evaluable Subjects with GP Assessment of BPH="Yes" and Urologist Assessment of BPH="No"
- Evaluable Subjects with GP Assessment of BPH="Yes" and Any Urologist Risk Assessment of BPH Progression
- Evaluable Subjects with GP Assessment of BPH="Yes" and Urologist Risk Assessment of BPH Progression="Yes"
- Evaluable Subjects with GP Assessment of BPH="Yes" and Urologist Risk Assessment of BPH Progression="No"

Serum PSA values will be presented by the following categories: IPSS\geq 8, BPE/BPO\geq 3, IPSS\geq 8 and BPE/BPO\geq 3, and IPSS\geq 8 or BPE/BPO\geq 3. The serum PSA data will also be presented by country, and separately by country and center.

A listing of the serum PSA data will be provided.

## 8.2.7. Digital Rectal Examinations

A digital rectal examination (DRE) is scheduled to be performed at Visit 3 and may be performed at the screening visit (Visit 1). The results of normal versus focal abnormality, in addition to clinical significance, will be summarized for each visit using the following categories: IPSS\geq 8, BPE/BPO\geq 3, IPSS\geq 8 and BPE/BPO\geq 3, and IPSS\geq 8 or BPE/BPO\geq 3. The digital rectal examination data will also be presented by country, and separately by country and center.

A listing of digital rectal examination data will be provided.

## 8.3. Pharmacokinetic Analyses

Pharmacokinetic (PK) samples were not collected. No PK analyses are planned for this study.

## 8.4. Pharmacodynamic (and / or Biomarker) Analyses

Pharmacodynamic and Biomarker samples were not collected. No pharmacodynamic or biomarker analyses are planned for this study.

# 8.5. Pharmacokinetic / Pharmacodynamic Analyses

Pharmacokinetic/pharmacodynamic samples were not collected. No pharmacokinetic/pharmacodynamic analyses are planned for this study.

#### 9. OTHER STATISTICAL ANALYSES

No other statistical analyses are planned for this study.
## 10. REFERENCES

GlaxoSmithKline Document Number 2012N140248\_02 Study ID FDC116114. Implementation of a screening tool for subjects with benign prostatic enlargement/obstruction to identify men ≥50 years presenting in General Practice with other co-morbidities who should be assessed for BPH. Effective Date 18Jan2016.

GlaxoSmithKline Document: Program Safety Analysis Plan (PSAP) for GI198745 (dutasteride) and GSK2285985 (fixed dose combination of dutasteride [GI198745] and tamsulosin [GI138525]); PSAP approval date 09Dec2016.

Landis, J.R.; Koch, G.G. The measurement of observer agreement for categorical data. *Biometrics*. 1977;33 (1): 159-174

Stokes, Maura E., Charles S. Davis, and Gary G. Koch. 2000. *Categorical Data Analysis Using the SAS® System, Second Edition*. Cary, NC: SAS Institute Inc.

# 11. APPENDICES

| Section | Appendix |
|---|---|
| RAP Section 4 | : Analysis Populations |
| Section 11.1 | Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population |
| RAP Section 5 | : Considerations for Data Analyses & Data Handling Conventions |
| Section 11.2 | Appendix 2: Time and Events |
| Section 11.3 | Appendix 3: Assessment Windows |
| Section 11.4 | Appendix 4: Treatment States & Phases |
| Section 11.5 | Appendix 5: Data Display Standards & Handling Conventions |
| | Study Treatment & Sub-group Display Descriptors |
| | Baseline Definitions & Derivations |
| | Reporting Process & Standards |
| Section 11.6 | Appendix 6: Derived and Transformed Data |
| | General |
| | Study Population |
| Section 11.7 | Appendix 7: Premature Withdrawals & Handling of Missing Data |
| | Premature Withdrawals |
| | Handling of Missing Data |
| | Handling of Missing Dates |
| | Handling of Partial Dates |
| Section 11.8 | Appendix 8: Adverse Event Time Periods and Special Adverse Event Definitions |
| Section 11.9 | Appendix 9: Values of Potential Clinical Importance |
| Section 11.10 | Appendix 10: Multicenter Studies |
| Section 11.11 | Appendix 11: Examination of Covariates, Subgroups, and Other Strata |
| Section 11.12 | Appendix 12: Multiple Comparisons and Multiplicity |
| Section 11.13 | Appendix 13: Model Checking and Diagnostics for Statistical Analyses |
| Other RAP App | endices |
| Section 11.14 | Appendix 14: Abbreviations & Trade Marks |
| Section 11.15 | Appendix 15: List of Data Displays |
| Section 11.16 | Appendix 16: Example Mock Shells for Data Displays |
| Section 11.17 | Appendix 17: Amendment 01 Revisions |

# 11.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population

#### 11.1.1. Exclusions from Per Protocol Population

No investigational study drug is being administered during this study.

This is a non-randomized, interventional study utilizing a questionnaire-based assessment of men in general practice, therefore the populations are not defined in the traditional sense; there will be no Per Protocol population for this study. The analysis population will be All Evaluable Subjects.

In accordance with SOP-130050 and the FDC116114 Protocol Deviation Management Plan (PDMP), a final review of the study deviations will be conducted by members of the internal and external Data Management team in advance of database freeze (DBF).

Below is a list of the deviations which are considered important as per the PDMP and will be summarized in a table by category; a supportive 'by subject' data listing will also be provided.

### Deviation Category:

be marked "IMP=N."

Informed Consent
Violation of Inclusion Criteria (Inclusion #)
Violation of Exclusion Criteria (Exclusion #)
Not Withdrawn After Developing Withdrawal Criteria
Excluded Medication, Vaccine, or Device
Assessment or Time Point Completion<sup>1</sup>

Failure to Report Safety Events per Protocol

<sup>1</sup> Deviations pertaining to incomplete and out of window assessments will be reviewed in-stream and assigned importance status during protocol deviation review meetings. Deviations related to missed assessments affecting subject safety will be marked "IMP = Y," deviations not affecting subject safety will

# 11.2. Appendix 2: Time & Events

## 11.2.1. Protocol Defined Time & Events

| Procedure | VISIT 1:<br>Screening/<br>Enrollment at GP Clinic | Study Period (1 week ±4 days to 6 weeks) | |
|---|---|---|---|
| Trocedure | | VISIT 2 (phone call):<br>GP | VISIT 3: Urologist <sup>6</sup><br>(up to 6 weeks after V1) |
| Informed consent | X | | |
| Inclusion and exclusion criteria | X | | |
| Demography | X | | |
| Medical history | X | | |
| Concomitant medications (all ongoing and within 30 days prior to Visit 1) | Х | | |
| IPSS screening tool | X | | |
| BPE/BPO screening tool | X | | |
| PROCEDURES AFTER SUBJECT IS ENROLLED <sup>1</sup> : | | | |
| Urine strip test <sup>2</sup> | Х | | |
| Urinalysis (only if urine strip test is positive) <sup>2</sup> | X | | |
| PSA blood test <sup>3</sup> | X | | |
| Results phone call to subject <sup>4</sup> | | X | |
| Digital rectal exam (DRE) <sup>5</sup> | X | | X |
| Brief physical examination | | | X |
| Enter prostate-related results in the CRF from non-protocol required procedures | | | Х |
| AE/SAE review (related to study procedures and/or participation) | <del>-=======</del> | <br>:==================================== | <u> </u><br>===== <del>-</del> |
| Concomitant medication review | <b>←=====</b> | | =====> |

- 1. Subject is enrolled after meeting eligibility requirements, which includes a positive BPE/BPO screening tool and/or positive IPSS screening tool.
- 2. Urinalysis sent to local laboratory only if urine strip test is positive.
- 3. PSA blood test sent to local lab. Local lab results and reference ranges are entered in the CRF.
- 4. For Visit 2, the GP calls the subject to report yes or no for probable BPH. If the subject has probable BPH, the GP schedules the subject for Visit 3 with the Urologist. If the subject does not have probable BPH, then the subject has completed the study.
- 5. DRE is performed by the Urologist. The GP may conduct a DRE at visit 1 however the DRE will be repeated by the Urologist to confirm the diagnosis and to rule out an abnormality suggesting prostate cancer.
- 6. Information collected during visit 3 will be entered into the eCRF by the Principal Investigator.

# 11.3. Appendix 3: Assessment Windows

No assessment windows for the statistical analysis are defined. If a subject is eligible for enrollment, diagnostic testing is performed at Visit 1.Visit 2 is a phone call from the GP to the subject within 1 week  $\pm$  4 days of Visit 1 detailing the diagnostic test results and a determination of probable BPH. Visit 3 is an Urologist assessment and should be completed within 6 weeks of Visit 1.

# 11.4. Appendix 4: Treatment States and Phases

There are no treatment states or phases for this study.

# 11.5. Appendix 5: Data Display Standards & Handling Conventions

#### 11.5.1. Study Treatment & Sub-group Display Descriptors

There are no study treatments for this study. However, results for IPSS and BPE/BPO screening tests will be displayed using the following groupings: IPSS≥8, BPE/BPO≥3, IPSS≥8 and BPE/BPO≥3, and IPSS≥8 or BPE/BPO≥3.

#### 11.5.2. Baseline Definition & Derivations

Baseline data are collected at Visit 1. No change from baseline values are calculated.

#### 11.5.3. Reporting Process & Standards

| Reporting Process | Reporting Process |
|---|---|
| Software | Software |
| software version | <ul> <li>SAS software will be used for all analyses except when noted. It is anticipated that the SAS software version 9.3 will be in use at statistical analysis complete; use of a version other than 9.3 will be documented in IMMS Study File.</li> </ul> |
| | e following server and areas are identified as of RAP finalization. Revisions to platform / server relocation, will be documented in IMMS Study File. |
| HARP Server | US1SALX00259 |
| HARP Area | The high level area is defined as: /arenv/arprod/gsk2285985/fdc116114/final. |
| QC Spreadsheet | QC process and documentation for analysis and reporting will be maintained as a text file on HARP server US1SALX00259 within above noted area. |
| Analysis Datasets | |
| Analysis datasets will be created according to Legacy GSK A&R dataset | |
| Generation of RTF Files | |
| | RTF files will be generated for all tabular summaries with the reporting efforts described in the RAP unless clearly stated as not required by the assigned Scientific and Medical Writer(s). |

#### **Reporting Standards**

#### General

The current GSK Integrated Data Standards Library (IDSL) and GSK IDSL Statistical Principles will be applied for reporting, unless otherwise stated within RAP text or indicated in table, listing, figure shells:

- 4.03 to 4.24: General Principles
- 5.01 to 5.08: Principles Related to Data Listings
- 6.01 to 6.11: Principles Related to Summary Tables
- 7.01 to 7.13: Principles Related to Graphics

From the above standards and principles as well as to be aligned with historical reporting for this

#### **Reporting Standards**

indication, the key reporting standards to be applied are:

- Within listings, numeric data will be reported at the precision collected in the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of decimal places.
- Within tabular summaries, the minimum and maximum values are presented with the same number of decimal places as the raw data collected on the eCRF. The mean and percentiles (e.g. median, Q1, and Q3) are presented using one additional decimal place. The standard deviation and standard error are presented using two additional decimal places.
- Continuous variables (e.g., age) will be summarized using the number of observations (n), mean, standard deviation (SD), median, minimum, and maximum.
- Categorical variables will be summarized using the number of subjects (n) and percentage (%) in each category.

#### **Planned and Actual Time**

- Reporting for tables, figures, data listings, and formal statistical analyses:
  - No investigational study drug is being administered during this study, therefore, there are no protocol-defined time windows.

#### **Unscheduled Visits**

There should be no unscheduled visits on this study.

#### **Descriptive Summary Statistics**

| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
|--------------------|--------------------------------------------|
| Categorical Data | N, n, frequency, % |
| Graphical Dieplaye | |

#### **Graphical Displays**

• Refer to IDSL Statistical Principals 7.01 to 7.13.

### 11.6. Appendix 6: Derived and Transformed Data

#### 11.6.1. **General**

No investigational study drug is being administered during this study. No data are transformed.

#### Date of Enrollment

An Evaluable Subject is a subject that was not a screen failure and also met the IPSS and/or BPE/BPO entry criteria (IPSS ≥8 and/or BPE/BPO ≥3). The Date of Enrollment is the later of the Screening date and IPSS and BPE/BPO assessment completion dates.

Study Day is calculated as the number of days from the Date of Enrollment:

- Enrollment Date = Missing → Study Day = Missing
- Reference Date < Enrollment Date → Study Day = Reference Date Enrollment Date
- Reference Date ≥ Enrollment Date → Study Day = Reference Date (Enrollment Date) + 1

#### 11.6.2. Study Population

#### **Demographics**

#### Age

Only year of birth is collected in the eCRF. For purposes of calculating age for a given subject, date of birth will be defined as June 30th of the corresponding year of birth. Age is calculated in terms of Screening (Visit 1) date and output as a truncated integer. Age categories include <65, ≥65, <75, ≥75 years.

#### Race

Race will be determined based on a subject's reported geographic ancestry as defined in the following table. Race information will not be presented for subjects who were enrolled in the study in France.

| Race | | | |
|---|---|---|---|
| | Asian | White | Other |
| Geographic | Any combination of<br>(restricted to the<br>categories below<br>only): | Any combination of<br>(restricted to the below<br>categories only) -White – Arabic/North | African American/African Heritage American Indian |
| Ancestry | -Asian – East Asian<br>Heritage | African Heritage<br>-White – | or Alaskan<br>Native |
| | -Asian – Japanese<br>Heritage | White/Caucasian/European<br>Heritage | Native Hawaiian<br>or Other Pacific<br>Islander |
| | -Asian – South<br>East Asian<br>Heritage | | |
| | -Asian – Central /<br>South Asian<br>Heritage | | |

## **Diagnostic Tests and Questionnaires**

IPSS (total score)

IPSS (total score) = Sum of IPSS individual questions 1-7.

BPE/BPO (total score)

BPE/BPO (total score) = Sum of BPE/BPO individual questions 1-3.

# 11.7. Appendix 7: Premature Withdrawals & Handling of Missing Data

## 11.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | Subject study completion (i.e. as specified in the protocol) was defined as completing Visits 1, 2, and 3. |
| | Withdrawn subjects were not replaced in the study. |
| | All available data from subjects who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified. |
| | Number and percent of Evaluable subjects completing the study and those withdrawing from the study, along with eCRF recorded reasons for premature withdrawals, will be summarized. |

## 11.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>No investigational study drug is being administered during this study.</li> <li>Subjects are not randomized or dispensed study treatment. As designed in the protocol, the number of subjects will decrease from the screening period to GP Assessment (Part II) and then again in the subsequent Urologist Assessment (Part III) either due to not qualifying for progression to the next part of the study or due to any withdrawal.</li> <li>The decreases, along with planned multiple summary and analysis types, will impact and restrict the evaluable population for a given endpoint. Therefore, populations are not defined in the traditional sense. There are no ITT or Per Protocol populations in this study. The analysis population will be All Evaluable Subjects.</li> <li>Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: <ul> <li>These data will be indicated by the use of a "blank" in subject listing displays. Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> <li>Answers such as "Not applicable" and "Not evaluable" or "Not Done" are not considered to be missing data and should be displayed as such.</li> <li>Due to the design of the study and types of endpoints incorporated, 'observed cases' will be summarized. For the primary analyses, there will be no imputations for missing data, no imputations for missing responses within the BPE/BPO or IPSS screening tools, and no imputations for subjects withdrawing from the study or not qualifying for a subsequent part of the study.</li> </ul> </li> </ul> |
| Outliers | Any subjects excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

# 11.7.2.1. Handling of Missing Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Adverse<br>Events | <ul> <li>The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: <ul> <li>Missing Start Day: First of the month will be used unless this is before the start date of the study; in this case the study start date will be used.</li> <li>Missing Stop Day: Last day of the month will be used, unless this is after the stop date of the study; in this case the study stop date will be used.</li> </ul> </li> </ul> |
| | <ul> <li>Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing.</li> <li>Start or end dates which are completely missing (i.e. no year specified) will remain missing, with no imputation applied.</li> </ul> |

# 11.7.2.2. Handling of Partial Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Concomitant<br>Medications | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> </li> <li>The recorded partial date will be displayed in listings.</li> </ul> |
| Adverse<br>Events | <ul> <li>Any partial dates for adverse events will be raised to data management. If the full date cannot be ascertained, the following assumptions will be made: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month.</li> <li>However, if this results in a date prior to Week 1 Day 1 and the event could possibly have occurred while on study from the partial information, then the Week 1 Day 1 date will be assumed to be the start date.</li> <li>The AE will then be considered to start on-study (worst case).</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> </li> <li>The recorded partial date will be displayed in listings.</li> </ul> |

# 11.8. Appendix 8: Adverse Event Time Periods and Special Adverse Event Definitions

Date-related derivations and transformations related to adverse events (AEs) are described below.

AE Onset Time since Enrollment

- = AE Onset Date Enrollment Date if Enrollment start date > AE onset date
- = AE Onset Date Enrollment Start Date +1 if Enrollment start date <= AE start date
- = missing otherwise

AE Duration (in days) = AE Resolution Date - AE Onset Date + 1

If the AE onset date is partially missing, the timing is determined as follows:

- 1. If the non-missing parts of the date (either just year or year/month) are unambiguously before the start of enrollment, the AE is considered Pre-Enrollment.
- 2. If the non-missing parts of the date are unambiguously after Visit 3, the AE is considered post-study.
- 3. If #1 or #2 above cannot be assigned, then the AE is considered during the study.

For computing AE duration, partial AE start and end dates will be imputed as previously described, and events with completely unknown (missing) end dates will be censored at the latter of the following two dates: date of last clinic visit, latest AE start date. AE duration is the total number of non-overlapping days for all events per subject, and will be considered censored if any contributing event is censored.

Time to death is defined as (date of death – enrollment date +1). For subjects who do not experience death, time to death is censored at the date of last clinic visit (if missing, the subject will be censored at the enrollment start date).

Special interest adverse events, including MedDRA preferred terms (MedDRA Version 19.1) and codes, are presented below in Tables A-D:

Table A: Sexual and Breast Adverse Events of Special Interest

Table B: Prostate Cancer Adverse Events of Special Interest

Table C: Cardiovascular Adverse Events of Special Interest

Table D: Infrequent Tier 1 Adverse Events of Special Interest

| Table A Sexual and Breast Adverse Events of Special Interest: MedDRA Preferred Terms and Codes | | |
|---|---|---|
| Special Interest Event | MedDRA Preferred Term | PT_Code |
| • | Sexual dysfunction | 10040477 |
| Altered (Decreased) Libido | Male sexual dysfunction | 10057672 |
| | Libido decreased | 10024419 |
| | Loss of libido | 10024870 |
| | Libido disorder | 10061221 |
| | Erectile dysfunction | 10061461 |
| Impotence | Organic erectile dysfunction | 10052004 |
| | Disturbance in sexual arousal | 10058929 |
| | Psychogenic erectile dysfunction | 10052005 |
| | Ejaculation delayed | 10014325 |
| Ejaculation Disorders | Ejaculation disorder | 10014326 |
| | Ejaculation failure | 10014328 |
| | Retrograde ejaculation | 10038967 |
| | Anorgasmia | 10002652 |
| | Orgasm abnormal | 10031085 |
| | Premature ejaculation | 10036596 |
| | Male orgasmic disorder | 10025513 |
| | Orgasmic sensation decreased | 10052449 |
| | Semen volume decreased | 10039944 |
| | Breast hyperplasia | 10006256 |
| Breast Disorders | Breast enlargement | 10006242 |
| | Gynaecomastia | 10018800 |
| | Nipple disorder | 10029417 |
| | Breast engorgement | 10006240 |
| | Breast swelling | 10006312 |
| | Breast pain | 10006298 |
| | Breast tenderness | 10006313 |
| | Nipple pain | 10029421 |
| | Nipple swelling | 10058680 |
| | Breast discomfort | 10049872 |
| | Breast hyperplasia | 10006256 |
| Breast Disorders: Breast Enlargement | Breast enlargement | 10006242 |
| | Gynaecomastia | 10018800 |
| | Nipple disorder | 10029417 |
| | Breast engorgement | 10006240 |
| | Breast swelling | 10006312 |
| | Breast pain | 10006298 |
| Breast Disorders: Breast Tenderness | Breast tenderness | 10006313 |
| | Nipple pain | 10029421 |
| | Nipple swelling | 10058680 |
| | Breast discomfort | 10049872 |

| Table B. Prostate Cancer Adverse Events of Special Interest: MedDRA Preferred Terms and Codes | | |
|---|---|---|
| Special Interest Event | Special Interest Event MedDRA Preferred Term PT_Code | |
| | Prostate cancer | 10060862 |
| | Prostate cancer stage 0 | 10036912 |
| Prostate Cancer | Prostate cancer stage I | 10036917 |
| | Prostate cancer stage II | 10036918 |
| | Prostate cancer stage III | 10036919 |
| | Prostate cancer stage IV | 10036920 |
| | Prostate cancer recurrent | 10036911 |
| | Prostate cancer metastatic | 10036909 |

| Table C. Cardiovascular Adverse Events of Special Interest: MedDRA Preferred Terms and Codes | | |
|---|---|---|
| Special Interest Event | MedDRA Preferred Term | PT_Code |
| | Acute myocardial infarction | 10000891 |
| | Myocardial infarction | 10028596 |
| Acute Coronary Syndrome | Silent myocardial infarction | 10049768 |
| | Sudden cardiac death | 10049418 |
| | Angina unstable | 10002388 |
| | Cardiac arrest | 10007515 |
| | Cardio-respiratory arrest | 10007617 |
| | Cardiac death | 10049993 |
| | Acute coronary syndrome | 10051592 |
| | Cerebrovascular accident | 10008190 |
| | Transient ischemic attack | 10044390 |
| Ischemic Cerebrovascular Events | Cerebral infarction | 10008118 |
| | Cerebrovascular disorder | 10008196 |
| | Cerebral artery embolism | 10008088 |
| | Cerebral artery occlusion | 10008089 |
| | Cerebral artery thrombosis | 10008092 |
| | Ischemic stroke | 10061256 |
| | Cerebral circulatory failure | 10008097 |
| | Cerebellar infarction | 10008034 |
| | Thalamic infarction | 10064961 |
| | Reversible ischemic neurologic deficit | 10050496 |
| | Thrombotic stroke | 10043647 |
| | Embolic stroke | 10014498 |
| | Vertebral artery occlusion | 10048965 |
| | Carotid arterial embolus | 10007684 |
| | Carotid artery occlusion | 10048964 |
| | Carotid artery stenosis | 10007687 |
| | Carotid artery thrombosis | 10007688 |
| | Thrombotic cerebral infarction | 10067347 |
| | Brain stem infarction | 10006147 |
| | Embolic cerebral infarction | 10060839 |
| | Lacunar infarction | 10051078 |
| | Brain stem stroke | 10068644 |
| | Stroke in evolution | 10059613 |
| | Ischaemic cerebral infarction | 10060840 |

| Table C Cardiovascular Adverse Events of Special Interest: MedDRA Preferred Terms and Codes (continued) | | |
|---|---|---|
| Special Interest Event | MedDRA Preferred Term | PT_Code |
| • | Cardiac failure congestive | 10007559 |
| | Cardiac failure | 10007554 |
| Cardiac Failure | Left ventricular failure | 10024119 |
| | Cardiac failure acute | 10007556 |
| | Cardiogenic shock | 10007625 |
| | Left ventricular failure acute | 10063081 |
| | Right ventricular failure | 10039163 |
| | Right ventricular failure acute | 10063082 |
| | Ventricular failure | 10060953 |
| | Cardiopulmonary failure | 10051093 |
| | Congestive cardiomyopathy | 10056370 |
| Ischemic Coronary Artery Disorders/ | Coronary artery embolism | 10011084 |
| Atherosclerosis | Coronary artery occlusion | 10011086 |
| | Coronary artery stenosis | 10011089 |
| | Coronary artery thrombosis | 10011091 |
| | Myocardial ischemia | 10028600 |
| | Coronary artery disease | 10011078 |
| | Arteriosclerosis coronary artery | 10003211 |
| | Ventricular extrasystoles | 10047289 |
| | Torsade de Pointes | 10044066 |
| Cardiac Arrhythmias | Ventricular fibrillation | 10047290 |
| | Cardiac Fibrillation | 10061592 |
| | Pulseless electrical activity | 10058151 |
| | Ventricular asystole | 10047284 |
| | Long QT syndrome | 10024803 |
| | Ventricular tachycardia | 10047302 |
| | Ventricular Arrhythmia | 10047281 |
| | Ventricular flutter | 10047294 |
| Peripheral Vascular Disease | Deep Vein Thrombosis | 10051055 |

| Table D. Infrequent Tier 1 Adverse Events of Special Interest: MedDRA Preferred Terms and Codes | | |
|---|---|---|
| Special Interest Event | MedDRA Preferred Term | PT_Code |
| Relevant for dutasteride: | | |
| | Anaphylactic reaction | 10002198 |
| | Anaphylactic shock | 10002199 |
| Allergic reactions | Anaphylactic transfusion reaction | 10067113 |
| | Anaphylactoid reaction | 10002216 |
| | Anaphylactoid shock | 10063119 |
| | Circulatory collapse | 10009192 |
| | Kounis syndrome | 10069167 |
| | Shock | 10040560 |
| | Type I hypersensitivity | 10045240 |
| | Allergic oedema | 10060934 |
| | Angioedema | 10002424 |
| | Circumoral oedema | 10052250 |
| | Conjunctival oedema | 10010726 |
| | Corneal oedema | 10011033 |
| | Epiglottic oedema | 10015029 |
| | Eye oedema | 10052139 |
| | Eye swelling | 10015967 |
| | Eyelid oedema | 10015993 |
| | Face oedema | 10016029 |
| | Gingival oedema | 10049305 |
| | Gingival swelling | 10018291 |
| | Gleich's syndrome | 10066837 |
| | Hereditary angioedema | 10019860 |
| | Idiopathic angioedema | 10073257 |
| | Idiopathic urticaria | 10021247 |
| | Laryngeal oedema | 10023845 |
| | Laryngotracheal oedema | 10023893 |
| | Limbal swelling | 10070492 |
| | Lip oedema | 10024558 |
| | Lip swelling | 10024570 |
| | Mouth Swelling | 10075203 |
| | Oculorespiratory syndrome | 10067317 |
| | Oedema mouth | 10030110 |
| | Oropharyngeal swelling | 10031118 |
| | Palatal oedema | 10056998 |
| | Palatal swelling | 10074403 |
| | Periorbital oedema | 10034545 |
| | Pharyngeal oedema | 10034829 |
| | Scleral oedema | 10057431 |
| | Swelling face | 10042682 |
| | Swollen tongue | 10042727 |
| | Tongue oedema | 10043967 |
| | Tracheal oedema | 10044296 |
| | Urticaria | 10046735 |
| | Urticaria cholinergic | 10046740 |
| | Urticaria chronic | 10052568 |
| | Urticaria papular | 10046750 |
| | Acquired epidermolysis bullosa | 10056508 |
| | Blister | 10005191 |
| | Blister rupture | 10073385 |
| | Bullous impetigo | 10006563 |

| Table D. Infrequent Tier 1 Adverse Ev and Codes | ents of Special Interest: MedDRA Prefer | red Terms |
|---|---|---|
| | Conjunctivitis | 10010741 |
| | Corneal exfoliation | 10064489 |
| | Drug eruption | 10013687 |
| | Epidermolysis | 10053177 |
| | Epidermolysis bullosa | 10014989 |
| | Genital ulceration | 10018180 |
| | HLA-B*1502 assay positive | 10074771 |
| | HLA-B*5801 assay positive | 10074774 |
| | Lip exfoliation | 10064482 |
| | Mouth ulceration | 10028034 |
| | Mucocutaneous ulceration | 10028084 |
| | Mucosa vesicle | 10028103 |
| | Mucosal erosion | 10061297 |
| | Mucosal exfoliation | 10064486 |
| | Mucosal necrosis | 10067993 |
| | Mucosal ulceration | 10028124 |
| | Nikolsky's sign | 10029415 |
| | Noninfective conjunctivitis | 10074701 |
| | Oral mucosal blistering | 10030995 |
| | Oral mucosal exfoliation | 10064487 |
| | Oral papule | 10031010 |
| | Oropharyngeal blistering | 10067950 |
| | Pemphigoid | 10034277 |
| | Pemphigus | 10034280 |
| | Penile exfoliation | 10064485 |
| | Skin erosion | 10040840 |
| | Skin exfoliation | 10040844 |
| | Staphylococcal scalded skin syndrome | 10041929 |
| | Stomatitis | 10042128 |
| | Tongue exfoliation | 10064488 |
| | Vaginal exfoliation | 10064483 |
| | Vaginal ulceration | 10046943 |
| | Vulval ulceration | 10047768 |
| | Vulvovaginal rash | 10071588 |
| | Vulvovaginal ulceration | 10050181 |
| | Application site pruritus | 10003053 |
| | Aquagenic pruritus | 10003071 |
| | Injection site pruritus | 10022093 |
| | Pruritus | 10037087 |
| | Pruritus genital | 10037093 |
| | Rash pruritic | 10037884 |
| | Senile pruritus | 10039986 |
| | Itching scar | 10050818 |
| | Eyelids pruritus | 10051627 |
| | Catheter site pruritus | 10052270 |
| | Pruritus generalised | 10052576 |
| | Infusion site pruritus | 10053664 |
| | Vulvovaginal pruritus | 10056530 |
| | Incision site pruritus | 10059386 |
| | Uraemic pruritus | 10060875 |
| | Pruritus allergic | 10063438 |
| | Instillation site pruritus | 10063763 |
| | Implant site pruritus | 10063785 |

| | Cholestatic pruritus | 10064190 |
|---|---|---|
| | Polymorphic eruption of pregnancy | 10066100 |
| | Vessel puncture site pruritus | 10067254 |
| | Vaccination site pruritus | 10067234 |
| | Brachioradial pruritus | 10071443 |
| | Notalgia paraesthetica | 10071443 |
| | Apocrine breast carcinoma | 10072043 |
| | Invasive breast carcinoma | 10000200 |
| Breast Cancer | Triple negative breast cancer | 10075715 |
| ricust Gariooi | Breast cancer | 10073300 |
| | Breast cancer female | 10057654 |
| | Breast cancer in situ | 10007034 |
| | Breast cancer male | 10061020 |
| | Breast cancer metastatic | 10051020 |
| | Breast cancer recurrent | 10003113 |
| | Breast cancer recurrent Breast cancer stage I | 10006198 |
| | Breast cancer stage II | 10006199 |
| | Breast cancer stage III | 10006200 |
| | Breast cancer stage IV | 10006201 |
| | Breast sarcoma | 10068582 |
| | Breast sarcoma metastatic | 10068583 |
| | Breast sarcoma recurrent | 10068584 |
| | Electron radiation therapy to breast | 10000304 |
| | Extended radical mastectomy | 10014437 |
| | Gamma radiation therapy to breast | 10013721 |
| | HER-2 positive breast cancer | 10065430 |
| | Inflammatory carcinoma of breast recurrent | 10021977 |
| | Inflammatory carcinoma of breast stage | 10021978 |
| | Inflammatory carcinoma of breast stage | 10021979 |
| | Inflammatory carcinoma of the breast | 10021980 |
| | Intraductal papillary breast neoplasm | 10073540 |
| | Intraductal proliferative breast lesion | 10073094 |
| | Invasive ductal breast carcinoma | 10073095 |
| | Invasive lobular breast carcinoma | 10073096 |
| | Invasive papillary breast carcinoma | 10073098 |
| | Lobular breast carcinoma in situ | 10073099 |
| | Malignant nipple neoplasm | 10062051 |
| | Malignant nipple neoplasm female | 10053129 |
| | Malignant nipple neoplasm male | 10053128 |
| | Mastectomy | 10026878 |
| | Medullary carcinoma of breast | 10027095 |
| | Medullary carcinoma of breast Metaplastic breast carcinoma | 10027095<br>10073100 |
| | Medullary carcinoma of breast Metaplastic breast carcinoma Modified radical mastectomy | 10027095<br>10073100<br>10027799 |
| | Medullary carcinoma of breast Metaplastic breast carcinoma Modified radical mastectomy Mucinous breast carcinoma | 10027095<br>10073100<br>10027799<br>10073101 |
| | Medullary carcinoma of breast Metaplastic breast carcinoma Modified radical mastectomy Mucinous breast carcinoma Neuroendocrine breast tumour | 10027095<br>10073100<br>10027799<br>10073101<br>10073103 |
| | Medullary carcinoma of breast Metaplastic breast carcinoma Modified radical mastectomy Mucinous breast carcinoma Neuroendocrine breast tumour Oestrogen receptor assay positive | 10027095<br>10073100<br>10027799<br>10073101 |
| | Medullary carcinoma of breast Metaplastic breast carcinoma Modified radical mastectomy Mucinous breast carcinoma Neuroendocrine breast tumour | 10027095<br>10073100<br>10027799<br>10073101<br>10073103 |

| and Codes | se Events of Special Interest: MedDRA Prefer | rieu rerms |
|---|---|---|
| | Photon radiation therapy to breast | 10034949 |
| | Postmastectomy lymphoedema | |
| | syndrome | 10036390 |
| | Progesterone receptor assay positive | 10054057 |
| | Radical mastectomy | 10037773 |
| | Radiotherapy to breast | 10062090 |
| | Simple mastectomy | 10040700 |
| | Tubular breast carcinoma | 10073104 |
| | X-ray therapy to breast | 10048199 |
| | Antioestrogen therapy | 10002816 |
| | Breast reconstruction | 10006305 |
| | Breast neoplasm | 10006279 |
| | Nipple neoplasm | 10056286 |
| | Phyllodes tumour | 10030280 |
| | Biopsy breast abnormal | 10071776 |
| | Breast calcifications | 10004745 |
| | Breast dysplasia | 10048782 |
| | | 10006237 |
| | Breast prosthesis implantation | 10006303 |
| | Computerised tomogram breast abnormal | 10074534 |
| | Activation syndrome | 10066817 |
| Depressed mood | Adjustment disorder with depressed | 122233.7 |
| - p | mood | 10001297 |
| | Columbia suicide severity rating scale | 1.200.201 |
| | abnormal | 10075616 |
| | Adjustment disorder with mixed anxiety | 1 2 2 2 3 2 . 0 |
| | and depressed mood | 10001299 |
| | Agitated depression | 10001496 |
| | Anhedonia | 10002511 |
| | Antidepressant therapy | 10054976 |
| | Childhood depression | 10068631 |
| | Decreased interest | 10011971 |
| | Depressed mood | 10012374 |
| | Depression | 10012378 |
| | Depression postoperative | 10012390 |
| | Depressive symptom | 10054089 |
| | Dysphoria | 10013954 |
| | Electroconvulsive therapy | 10014404 |
| | Feeling guilty | 10049708 |
| | Feeling of despair | 10016344 |
| | Feelings of worthlessness | 10016374 |
| | Major depression | 10057840 |
| | Menopausal depression | 10067371 |
| | Post stroke depression | 10070606 |
| | Postictal depression | 10070000 |
| | Completed suicide | 10011144 |
| | Depression suicidal | 10010144 |
| | Intentional overdose | 10012397 |
| | Intentional overdose | 10022524 |
| | Poisoning deliberate | 10022324 |
| | | 1 10000000 |
| | Self-injurious ideation | 10051154 |

| Table D. Infrequent Tier 1 Adverse Ev and Codes | ents of Special Interest: MedDRA Prefe | erred Terms |
|---|---|---|
| | Suicidal ideation | 10042458 |
| | Suicide attempt | 10042464 |
| | Alopecia | 10001760 |
| | Alopecia areata | 10001761 |
| Hair changes | Alopecia scarring | 10001764 |
| · · | Alopecia syphilitic | 10001765 |
| | Alopecia totalis | 10001766 |
| | Alopecia universalis | 10001767 |
| | Hypotrichosis | 10021126 |
| | Progeria | 10036794 |
| | Madarosis | 10051235 |
| | Follicular mucinosis | 10056506 |
| | Application site alopecia | 10059046 |
| | Androgenetic alopecia | 10068168 |
| | Satoyoshi syndrome | 10070579 |
| | Radiation alopecia | 10072045 |
| | Diffuse alopecia | 10072043 |
| | Hypertrichosis | 10020864 |
| | Congenital vas deferens absence | 10010670 |
| | Cryptorchism | 10010070 |
| Interference with formation of external | Epispadias | 10011498 |
| genitalia in a male fetus | Hypospadias | 10013008 |
| germana iri a maie retas | Reproductive tract hypoplasia, male | 10021093 |
| | Testicular dysplasia Congenital genital malformation male | 10059271<br>10059492 |
| | Penoscrotal fusion | 10059492 |
| | | 10064951 |
| | Sertoli-cell-only syndrome | 1006633 |
| | Buried penis syndrome | |
| | Penoscrotal transposition | 10067287 |
| | Penile torsion | 10070235 |
| | Infertility tests | 10021931 |
| Detential for decreased male fortility | pH semen | 10034784 |
| Potential for decreased male fertility | pH semen decreased | 10034786 |
| | pH semen increased | 10034788 |
| | pH semen normal | 10034790 |
| | Red blood cells semen | 10038176 |
| | Red blood cells semen negative | 10038179 |
| | Red blood cells semen positive | 10038180 |
| | Semen liquefaction | 10039931 |
| | Semen liquefaction normal | 10039933 |
| | Semen liquefaction prolonged | 10039934 |
| | Semen liquefaction shortened | 10039935 |
| | Semen viscosity | 10039936 |
| | Semen viscosity decreased | 10039938 |
| | Semen viscosity increased | 10039940 |
| | Semen viscosity normal | 10039942 |
| | Semen volume abnormal | 10039943 |
| | Semen volume decreased | 10039944 |
| | Semen volume increased | 10039946 |
| | Semen volume normal | 10039948 |
| | Sperm analysis | 10041476 |
| | Sperm analysis abnormal | 10041477 |
| | Sperm analysis normal | 10041478 |

| and Codes | Cnownoto | 10044400 |
|---|---|---|
| | Spermatozoa abnormal | 10041498 |
| | Spermatozoa morphology | 10041501 |
| | Spermatozoa morphology abnormal | 10041502 |
| | Spermatozoa morphology normal | 10041503 |
| | Spermatozoa progressive motility | 40044504 |
| | abnormal | 10041504 |
| | Spermatozoa progressive motility | 10011500 |
| | decreased | 10041506 |
| | Spermatozoa progressive motility | 10041507 |
| | normal | 10041507 |
| | White blood cells semen | 10047956 |
| | White blood cells semen negative | 10047959 |
| | White blood cells semen positive | 10047960 |
| | Fructose semen decreased | 10052476 |
| | Fructose semen increased | 10052477 |
| | Prostatic fluid leukocytes increased | 10053866 |
| | Infertility tests abnormal | 10062020 |
| | Infertility tests normal | 10062021 |
| | pH semen abnormal | 10062074 |
| | Semen liquefaction abnormal | 10062159 |
| | Semen viscosity abnormal | 10062160 |
| | Semen analysis normal | 10062238 |
| | Semen analysis | 10068482 |
| | Semen analysis abnormal | 10068483 |
| | Sperm concentration decreased | 10070925 |
| | Sperm concentration increased | 10070926 |
| | Sperm concentration abnormal | 10070927 |
| | Sperm concentration normal | 10070928 |
| | Sperm concentration | 10070929 |
| | Sperm concentration zero | 10070930 |
| | Total sperm count | 10070931 |
| | Total sperm count decreased | 10070932 |
| | Infertility | 10021926 |
| | Infertility male | 10021929 |
| | Anorchism | 10002641 |
| | Eunuchoidism | 10015532 |
| esticular pain and swelling | Hypogonadism male | 10021011 |
| | Testicular atrophy | 10043298 |
| | Testicular disorder | 10043306 |
| | Testicular failure | 10043315 |
| | Testicular failure postoperative | 10043317 |
| | Testicular failure primary | 10043318 |
| | Testicular hyperfunction | 10043334 |
| | Testicular infarction | 10043337 |
| | Testicular pain | 10043345 |
| | Testicular retraction | 10043348 |
| | Testicular swelling | 10043354 |
| | Testicular torsion | 10043356 |
| | Testicular necrosis | 10049572 |
| | Spermatic cord mass | 10049792 |
| | Testicular appendage torsion | 10050476 |
| | Spermatic cord pain | 10051221 |

| Table D. Infrequent Tier 1 Adverse<br>and Codes | Events of Special Interest: MedDRA Prefe | erred Terms |
|---|---|---|
| | Testicular injury | 10051872 |
| | Testicular haemorrhage | 10051877 |
| | Epididymal calculus | 10052321 |
| | Epididymal enlargement | 10052322 |
| | Epididymal tenderness | 10052323 |
| | Testis discomfort | 10052531 |
| | Monorchidism | 10055002 |
| | Epididymal disorder | 10055045 |
| | Spermatic cord disorder | 10056348 |
| | Testicular mass | 10058901 |
| | Testotoxicosis | 10063654 |
| | Spermatic cord haemorrhage | 10065742 |
| | Spermatic cord obstruction | 10065805 |
| | Spermatic cord perforation | 10065806 |
| | Spermatic cord stenosis | 10065807 |
| | Testicular perforation | 10065808 |
| | Testicular hypertrophy | 10066101 |
| | Testicular oedema | 10066769 |
| | Sperm granuloma | 10067802 |
| | Testicular microlithiasis | 10067829 |
| | Congenital monorchidism | 10069505 |
| | Testicular autoimmunity | 10071574 |
| Relevant for tamsulosin: | . sociodiai datomininti | 1007 107 4 |
| | Arrhythmia | 10003119 |
| Atrial fibrillation, tachycardia, | Heart alternation | 10058155 |
| arrhythmias | Heart rate irregular | 10019304 |
| | Pacemaker generated arrhythmia | 10053486 |
| | Pacemaker syndrome | 10051994 |
| | Paroxysmal arrhythmia | 10050106 |
| | Pulseless electrical activity | 10058151 |
| | Reperfusion arrhythmia | 10058156 |
| | Withdrawal arrhythmia | 10047997 |
| | Arrhythmia supraventricular | 10003130 |
| | Atrial fibrillation | 10003658 |
| | Atrial flutter | 10003662 |
| | Atrial parasystole | 10071666 |
| | Atrial tachycardia | 10003668 |
| | Junctional ectopic tachycardia | 10074640 |
| | Sinus tachycardia | 10040752 |
| | Supraventricular extrasystoles | 10042602 |
| | Supraventricular tachyarrhythmia | 10065342 |
| | Supraventricular tachycardia | 10042604 |
| | ECG P wave inverted | 10057526 |
| | Electrocardiogram P wave abnormal | 100573284 |
| | Retrograde p-waves | 10071187 |
| | Anomalous atrioventricular excitation | 10002611 |
| | Cardiac flutter | 10052840 |
| | Extrasystoles | 10032040 |
| | Tachyarrhythmia | 10013836 |
| | Accelerated idioventricular rhythm | 10049447 |
| | Cardiac fibrillation | 10049003 |
| | Parasystole | 10001392 |
| | <sub> </sub> 1 นานองอเบเซ | 1 10000022 |

| Table D. Infrequent Tier 1 Advers | se Events of Special Interest: MedDRA Prefe | erred Terms |
|---|---|---|
| | Torsade de pointes | 10044066 |
| | Ventricular arrhythmia | 10047281 |
| | Ventricular extrasystoles | 10047289 |
| | Ventricular fibrillation | 10047290 |
| | Ventricular flutter | 10047294 |
| | Ventricular parasystole | 10058184 |
| | Ventricular pre-excitation | 10049761 |
| | Ventricular tachyarrhythmia | 10065341 |
| | Ventricular tachycardia | 10047302 |
| Floppy Iris Syndrome | , | |
| | Floppy iris syndrome | 10066373 |
| | Dizziness | 10013573 |
| | Dizziness postural | 10013578 |
| Orthostasis | Orthostatic hypotension | 10031127 |
| | Hypotension | 10021097 |
| | Syncope | 10042772 |
| | Presyncope | 10036653 |
| | Blood pressure orthostatic abnormal | 10053354 |
| | Blood pressure orthostatic decreased | 10053356 |
| Priapism | Priapism | 10036661 |
| | Acute generalised exanthematous pustulosis | 10048799 |
| Stevens-Johnson syndrome | Cutaneous vasculitis | 10011686 |
| -<br>- | Dermatitis bullous | 10012441 |
| | Dermatitis exfoliative | 10012455 |
| | Dermatitis exfoliative generalised | 10012456 |
| | Drug reaction with eosinophilia and | |
| | systemic symptoms | 10073508 |
| | Epidermal necrosis | 10059284 |
| | Erythema multiforme | 10015218 |
| | Exfoliative rash | 10064579 |
| | Oculomucocutaneous syndrome | 10030081 |
| | Skin necrosis | 10040893 |
| | Stevens-Johnson syndrome | 10042033 |
| | Toxic epidermal necrolysis | 10044223 |
| | Toxic skin eruption | 10057970 |

# 11.9. Appendix 9: Values of Potential Clinical Importance

# 11.9.1. Laboratory Values

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (> x) |
| Prostate Specific Antigen (PSA) | Ng/mL | NA | Not Applicable | 9.9 |

| Urinalysis | | | |
|---|---|---|---|
| Test Analyte | Units | Category | Clinical Concern Range |
| Urine Dipstick | NA | Pos / Neg | Not Applicable |
| Urine Glucose (dipstick) | NA | Pos / Neg | Not Applicable |
| Urine Microscopy – Red Blood<br>Cells | NA | Pos / Neg | Not Applicable |
| Urine Leukocyte Esterase test for detecting WBC (dipstick) | NA | Pos / Neg | Not Applicable |
| Urine Protein (dipstick) | NA | Pos / Neg | Not Applicable |

# 11.10. Appendix 10: Multicenter Studies

## 11.10.1. Methods for Handling Centers

- The countries participating in this trial include: Russia, Germany, Italy, France, and Spain.
- In this multicentre study, enrollment will be presented by country, and separately by country and center.

# 11.11. Appendix 11: Examination of Covariates, Subgroups & Other Strata

## **11.11.1.** Subgroups

- Covariates and Other Strata will not be used to perform the analysis.
- The following subgroups may be used in descriptive summaries and statistical analyses:
  - Country
  - Center

# 11.12. Appendix 12: Multiple Comparisons & Multiplicity

## 11.12.1. Handling of Multiple Comparisons & Multiplicity

All pre-planned summary statistics results will be presented. There are no established controls for interpretation of the multiple outputs.

# 11.13. Appendix 13: Model Checking and Diagnostics for Statistical Analyses

No models were used during the statistical analysis; only proportions and confidence intervals were calculated.

# 11.14. Appendix 14: Abbreviations and Trademarks

## 11.14.1. Abbreviations

| AE | Adverse Event |
|--------|----------------------------------------------------------|
| ВРН | Benign prostatic hyperplasia |
| BPE | Benign prostatic enlargement |
| BPO | Benign prostatic obstruction |
| CSR | Clinical Study Report |
| eCRF | Electronic case report form |
| DRE | Digital rectal examination |
| GSK | GlaxoSmithKline |
| GP | General Practitioner |
| IPSS | International Prostate Symptom Score (Version 2), I-PSS2 |
| MedDRA | Medical Dictionary for Regulatory Activities |
| PD | Pharmacodynamic |
| PK | Pharmacokinetic |
| PSA | Prostate specific antigen |
| RAP | Reporting and analysis plan |
| SAE | Serious adverse event |

## 11.14.2. Trademarks

| Trademarks of the GlaxoSmithKline<br>Group of Companies |
|---------------------------------------------------------|
| NONE |

Trademarks not owned by the GlaxoSmithKline Group of Companies

# 11.15. Appendix 15: List of Data Displays

# 11.15.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|---------------------------------------|------------|
| Study Population | 1.1 to 1.29 | NA |
| Efficacy | 2.1 to 2.54 | 2.1 to 2.3 |
| Safety | 3.1 to 3.31 | NA |
| Section | List | ings |
| ICH Listings | 1.3-1.7, 1.10-1.11, 2.1, 2.3, 3.2-3.9 | |
| Other Listings | 1.1-1.2, 1.8-1.9, 2.2, 3.1, 3.10-3.12 | |

# 11.15.2. Study Population Tables

| Stud | Study Population Tables | |
|---|---|---|
| No | Population | Title |
| Рори | Population: All Screened Subjects | |
| 1.1. | All Screened Subjects | Summary of Subject Accountability for Screened Subjects |
| 1.2. | All Screened Subjects | Summary of Screened Subjects by Country |
| 1.3. | All Screened Subjects | Summary of Screened Subjects by Country and Center |
| Popu | ulation: Screened But N | ot Evaluable Subjects |
| 1.4. | Screened But Not<br>Evaluable Subjects | Summary of Demographic Characteristics for Subjects Who Were Screened But Not Evaluable |
| 1.5. | Screened But Not<br>Evaluable Subjects | Summary of Inclusion/Exclusion Criteria Deviations for Subjects Who Were Screened But Not Evaluable |
| Popu | ılation: All Evaluable S | ubjects |
| 1.6. | All Evaluable Subjects | Summary of Subject Accountability for Evaluable Subjects |
| 1.7. | All Evaluable Subjects | Summary of Subject Accountability for Evaluable Subjects by Country |
| 1.8. | All Evaluable Subjects | Summary of Subject Accountability for Evaluable Subjects by Country and Center |
| 1.9. | All Evaluable Subjects | Summary of Evaluable Subjects by Country |
| 1.10. | All Evaluable Subjects | Summary of Evaluable Subjects by Country and Center |
| 1.11. | All Evaluable Subjects | Summary of Subject Disposition |
| 1.12. | All Evaluable Subjects | Summary of Subject Discontinuation by Visit |
| 1.13. | All Evaluable Subjects | Summary of Primary Reason for Study Withdrawal, by Period of Discontinuation |
| 1.14. | All Evaluable Subjects | Summary of Important Protocol Deviations for Evaluable Subjects |
| 1.15. | 1.15 All Evaluable Subjects Summary of Demographic Characteristics for Evaluable Subjects | |
| 1.16 All Evaluable Subjects Summary of Demographic Characteristics for Evaluable Subjects by Country | | , , , |
| 1.17. | All Evaluable Subjects | Summary of Demographic Characteristics for Evaluable Subjects by Country and Center |
| 1.18. | All Evaluable Subjects | Summary of Race |
| 1.19. | All Evaluable Subjects | Summary of Race by Country |
| 1.20. | All Evaluable Subjects | Summary of Race by Country and Center |
| 1.21. | 1. All Evaluable Subjects Summary of PSA Values at Visit 1 | |
| 1.22. | .22 All Evaluable Subjects Summary of PSA Values at Visit 1 by Country | |
| 1.23. | 23 All Evaluable Subjects Summary of PSA Values at Visit 1 by Country and Center | |
| 1.24. | 24. All Evaluable Subjects Summary of BPE/BPO and IPSS at Visit 1 | |
| 1.25. | .25 All Evaluable Subjects Summary of BPE/BPO and IPSS at Visit 1 by Country | |
| 1.26. | 1.26 All Evaluable Subjects Summary of BPE/BPO and IPSS at Visit 1 by Country and Center | |
| 1.27. | All Evaluable Subjects | Summary of Specific Medical Conditions at Screening |

| Stud | Study Population Tables | |
|---|---|---|
| No Population Title | | Title |
| 1.28. | All Evaluable Subjects | Summary of Surgical/Diagnostic Procedures |
| 1.29. | All Evaluable Subjects | Summary of Concomitant Medications |

# 11.15.3. Efficacy Tables

| Effic | Efficacy: Tables | |
|---|---|---|
| No | Population | Title |
| Рори | ılation: All Screened Su | ubjects |
| 2.1. | All Screened Subjects | Summary of Agreement Between BPE/BPO and IPSS Screening Tools |
| 2.2. | All Screened Subjects | Summary of Agreement Between BPE/BPO and IPSS Screening Tools by Country |
| 2.3. | All Screened Subjects | Summary of Agreement Between BPE/BPO and IPSS Screening Tools by Country and Center |
| Popu | ılation: All Evaluable S | ubjects |
| 2.4. | All Evaluable Subjects | Summary of IPSS Scores at Visit 1 by Subgroup |
| 2.5. | All Evaluable Subjects | Summary of IPSS Scores at Visit 1 by Country and Subgroup |
| 2.6. | All Evaluable Subjects | Summary of IPSS Scores at Visit 1 by Country, Center, and Subgroup |
| 2.7. | All Evaluable Subjects | Summary of BPH-Related Health Status at Visit 1 (IPSS Question 8) |
| 2.8. | All Evaluable Subjects | Summary of BPH-Related Health Status at Visit 1 (IPSS Question 8) by Country |
| 2.9. | All Evaluable Subjects | Summary of BPH-Related Health Status at Visit 1 (IPSS Question 8) by Country and Center |
| 2.10. | All Evaluable Subjects | Summary of BPE/BPO Scores at Visit 1 by Subgroup |
| 2.11. | All Evaluable Subjects | Summary of BPE/BPO Scores at Visit 1 by Country and Subgroup |
| 2.12. | All Evaluable Subjects | Summary of BPE/BPO Scores at Visit 1 by Country, Center, and Subgroup |
| 2.13. | All Evaluable Subjects | Summary of BPH Diagnosis by Urologist Based Upon BPE/BPO Score (≥3) |
| 2.14. | All Evaluable Subjects | Summary of BPH Diagnosis by Urologist Based Upon BPE/BPO Score (≥3) by Country |
| 2.15. | All Evaluable Subjects | Summary of BPH Diagnosis by Urologist Based Upon BPE/BPO Score (≥3) by Country and Center |
| 2.16. | All Evaluable Subjects | Summary of BPH Diagnosis by Urologist Based Upon IPSS Score (≥8) |
| 2.17. | All Evaluable Subjects | Summary of BPH Diagnosis by Urologist Based Upon IPSS Score (≥8) by Country |
| 2.18. | All Evaluable Subjects | Summary of BPH Diagnosis by Urologist Based Upon IPSS Score (≥8) by Country and Center |
| 2.19. | All Evaluable Subjects | Summary of BPH Diagnosis by Urologist Based Upon IPSS Score (≥8) or BPE/BPO Score (≥3) |
| 2.20. | All Evaluable Subjects | Summary of BPH Diagnosis by Urologist Based Upon IPSS Score (≥8) or BPE/BPO Score (≥3) by Country |
| 2.21. | All Evaluable Subjects | Summary of BPH Diagnosis by Urologist Based Upon IPSS Score (≥8) or BPE/BPO Score (≥3) by Country and Center |
| 2.22. | All Evaluable Subjects | Summary of BPH Diagnosis by Urologist Based Upon IPSS Score (≥8) and BPE/BPO Score (≥3) |

| Effic | Efficacy: Tables | |
|---|---|---|
| No | Population | Title |
| 2.23. | All Evaluable Subjects | Summary of BPH Diagnosis by Urologist Based Upon IPSS Score (≥8) and BPE/BPO Score (≥3) by Country |
| 2.24. | All Evaluable Subjects | Summary of BPH Diagnosis by Urologist Based Upon IPSS Score (≥8) and BPE/BPO Score (≥3) by Country and Center |
| 2.25. | All Evaluable Subjects | Summary of BPH Progression Risk by Urologist Based Upon BPE/BPO Score (≥3) |
| 2.26. | All Evaluable Subjects | Summary of BPH Progression Risk by Urologist Based Upon BPE/BPO Score (≥3) by Country |
| 2.27. | All Evaluable Subjects | Summary of BPH Progression Risk by Urologist Based Upon BPE/BPO Score (≥3) by Country and Center |
| 2.28. | All Evaluable Subjects | Summary of BPH Progression Risk by Urologist Based Upon IPSS Score (≥8) |
| 2.29. | All Evaluable Subjects | Summary of BPH Progression Risk by Urologist Based Upon IPSS Score (≥8) by Country |
| 2.30. | All Evaluable Subjects | Summary of BPH Progression Risk by Urologist Based Upon IPSS Score (≥8) by Country and Center |
| 2.31. | All Evaluable Subjects | Summary of BPH Progression Risk by Urologist Based Upon IPSS Score (≥8) or BPE/BPO Score (≥3) |
| 2.32. | All Evaluable Subjects | Summary of BPH Progression Risk by Urologist Based Upon IPSS Score (≥8) or BPE/BPO Score (≥3) by Country |
| 2.33. | All Evaluable Subjects | Summary of BPH Progression Risk by Urologist Based Upon IPSS Score (≥8) or BPE/BPO Score (≥3) by Country and Center |
| 2.34. | All Evaluable Subjects | Summary of BPH Progression Risk by Urologist Based Upon IPSS Score (≥8) and BPE/BPO Score (≥3) |
| 2.35. | All Evaluable Subjects | Summary of BPH Progression Risk by Urologist Based Upon IPSS Score (≥8) and BPE/BPO Score (≥3) by Country |
| 2.36. | All Evaluable Subjects | Summary of BPH Progression Risk by Urologist Based Upon IPSS Score (≥8) and BPE/BPO Score (≥3) by Country and Center |
| 2.37. | All Evaluable Subjects | Summary of Probable BPH Diagnosis by GP Based Upon BPE/BPO Score (≥3) |
| 2.38. | All Evaluable Subjects | Summary of Probable BPH Diagnosis by GP Based Upon BPE/BPO Score (≥3) by Country |
| 2.39. | All Evaluable Subjects | Summary of Probable BPH Diagnosis by GP Based Upon BPE/BPO Score (≥3) by Country and Center |
| 2.40. | All Evaluable Subjects | Summary of Probable BPH Diagnosis by GP Based Upon IPSS Score (≥8) |
| 2.41. | All Evaluable Subjects | Summary of Probable BPH Diagnosis by GP Based Upon IPSS Score (≥8) by Country |
| 2.42. | All Evaluable Subjects | Summary of Probable BPH Diagnosis by GP Based Upon IPSS Score (≥8) by Country and Center |
| 2.43. | All Evaluable Subjects | Summary of Probable BPH Diagnosis by GP Based Upon IPSS Score (≥8) or BPE/BPO Score (≥3) |

| Effic | Efficacy: Tables | |
|---|---|---|
| No | Population | Title |
| 2.44. | All Evaluable Subjects | Summary of Probable BPH Diagnosis by GP Based Upon IPSS Score (≥8) or BPE/BPO Score (≥3) by Country |
| 2.45. | All Evaluable Subjects | Summary of Probable BPH Diagnosis by GP Based Upon IPSS Score (≥8) or BPE/BPO Score (≥3) by Country and Center |
| 2.46. | All Evaluable Subjects | Summary of Probable BPH Diagnosis by GP Based Upon IPSS Score (≥8) and BPE/BPO Score (≥3) |
| 2.47. | All Evaluable Subjects | Summary of Probable BPH Diagnosis by GP Based Upon IPSS Score (≥8) and BPE/BPO Score (≥3) by Country |
| 2.48. | All Evaluable Subjects | Summary of Probable BPH Diagnosis by GP Based Upon IPSS Score (≥8) and BPE/BPO Score (≥3) by Country and Center |
| 2.49. | All Evaluable Subjects | Summary of Subjects Who Discontinued From the Study Before the GP Was Able to Assess the Presence of Probable BPH |
| 2.50. | All Evaluable Subjects | Summary of Subjects Who Discontinued From the Study Before the GP Was Able to Assess the Presence of Probable BPH by Country |
| 2.51. | All Evaluable Subjects | Summary of Subjects Who Discontinued From the Study Before the GP Was Able to Assess the Presence of Probable BPH by Country and Center |
| 2.52. | All Evaluable Subjects | Summary of Subjects Who Withdrew From the Study Before a Urologist Visit, Among Subjects Who Were Eligible for Such a Visit |
| 2.53. | All Evaluable Subjects | Summary of Subjects Who Withdrew From the Study Before a Urologist Visit, Among Subjects Who Were Eligible for Such a Visit by Country |
| 2.54. | All Evaluable Subjects | Summary of Subjects Who Withdrew From the Study Before a Urologist Visit, Among Subjects Who Were Eligible for Such a Visit by Country and Center |

# 11.15.4. Efficacy Figures

| Effic | Efficacy: Figures | |
|---|---|---|
| No | Population | Title |
| Popu | Population: All Evaluable Subjects | |
| 2.1. | All Evaluable<br>Subjects | Plot of IPSS Scores Versus BPE/BPO Scores at Visit 1 for All Evaluable Subjects |
| 2.2. | All Evaluable<br>Subjects | Plot of IPSS Scores Versus PSA Values at Visit 1 for All Evaluable Subjects |
| 2.3. | All Evaluable<br>Subjects | Plot of BPE/BPO Scores Versus PSA Values at Visit 1 for All Evaluable Subjects |

# 11.15.5. Safety Tables

| Safe | Safety : Tables | |
|---|---|---|
| No | Population | Title |
| Popu | ulation: All Evaluable S | ubjects |
| 3.1. | All Evaluable Subjects | Summary of Adverse Events by Type Starting Post-Enrollment |
| 3.2. | All Evaluable Subjects | Summary of Adverse Events Starting Post-Enrollment |
| 3.3. | All Evaluable Subjects | Summary of Non-Serious Adverse Events Starting Post-Enrollment |
| 3.4. | All Evaluable Subjects | Summary of Adverse Events Starting Post-Enrollment by Age Group (<65, ≥65) |
| 3.5. | All Evaluable Subjects | Summary of Adverse Events Starting Post-Enrollment by Age Group (<75, ≥75) |
| 3.6. | All Evaluable Subjects | Summary of Adverse Events Starting Post-Enrollment by Country |
| 3.7. | All Evaluable Subjects | Summary of Adverse Events Starting Post-Enrollment by Country and Center |
| 3.8. | All Evaluable Subjects | Summary of Adverse Events Starting post-Enrollment by Maximum Intensity |
| 3.9. | All Evaluable Subjects | Summary of Most Common Adverse Events Starting Post-Enrollment |
| 3.10. | All Evaluable Subjects | Summary of Most Common Non-Serious Adverse Events Starting Post-<br>Enrollment |
| 3.11. | All Evaluable Subjects | Summary of Serious Adverse Events Starting Post-Enrollment |
| 3.12. | All Evaluable Subjects | Summary of Serious Adverse Events Starting Post-Enrollment by Age Group (<65, ≥65) |
| 3.13. | All Evaluable Subjects | Summary of Serious Adverse Events Starting Post-Enrollment by Age Group (<75, ≥75) |
| 3.14. | All Evaluable Subjects | Summary of Serious Adverse Events Starting Post-Enrollment by Country |
| 3.15. | All Evaluable Subjects | Summary of Serious Adverse Events Starting Post-Enrollment by Country and Center |
| 3.16. | All Evaluable Subjects | Summary of Fatal Adverse Events Starting Post-Enrollment |
| 3.17. | All Evaluable Subjects | Summary of Adverse Events Starting Post-Enrollment Leading to Withdrawal From the Study |
| 3.18. | All Evaluable Subjects | Summary of Serious Adverse Events Starting Post-Enrollment Leading to Withdrawal From the Study |
| 3.19. | All Evaluable Subjects | Summary of Sexual and Breast Adverse Events of Special Interest Starting Post-Enrollment |
| 3.20. | All Evaluable Subjects | Summary of Special Interest Adverse Events Starting Post-Enrollment: Prostate Cancer |
| 3.21. | All Evaluable Subjects | Summary of Cardiovascular Adverse Events of Special Interest Starting Post-Enrollment |
| 3.22. | All Evaluable Subjects | Summary of Infrequent Tier I Special Interest Adverse Events Starting Post-<br>Enrollment |
| 3.23. | All Evaluable Subjects | Summary of PSA (ng/mL) at Visit 1 by Subgroup |

| Safe | Safety : Tables | |
|---|---|---|
| No | Population | Title |
| 3.24. | All Evaluable Subjects | Summary of PSA (ng/mL) at Visit 1 by Country and Subgroup |
| 3.25. | All Evaluable Subjects | Summary of PSA (ng/mL) at Visit 1 by Country, Center, and Subgroup |
| 3.26. | All Evaluable Subjects | Summary of Laboratory Data at Visit 1 |
| 3.27. | All Evaluable Subjects | Summary of Laboratory Data at Visit 1 by Country |
| 3.28. | All Evaluable Subjects | Summary of Laboratory Data at Visit 1 by Country and Center |
| 3.29. | All Evaluable Subjects | Summary of Digital Rectal Examination |
| 3.30. | All Evaluable Subjects | Summary of Digital Rectal Examination by Country |
| 3.31. | All Evaluable Subjects | Summary of Digital Rectal Examination by Country and Center |

## 11.15.6. ICH Listings

The following categorizes data listings as ICH (International Conference on Harmonization) used to support critical analyses or non-ICH. The two classifications are assigned with consideration for general regulatory requirements across countries at point of RAP finalization. Changes to these classifications may occur at point of reporting as a result of specific country requirements or requests and will not result in a RAP revision.

| ioii a | 1 | ICH Listings | |
|---|---|---|---|
| ICH | Non-<br>ICH | Study Population | Title |
| | 1.1 | Screened But Not<br>Evaluable | Listing of Demographic Characteristics for Subjects Who Were Screened But Not Evaluable |
| | 1.2 | Screened But Not<br>Evaluable | Listing of Subjects With Inclusion/Exclusion Criteria Deviations Who Were Screened But Not Evaluable |
| 1.3 | | All Evaluable Subjects | Listing of Subject Accountability |
| 1.4 | | All Evaluable Subjects | Listing of Reasons for Study Withdrawal |
| 1.5 | | All Evaluable Subjects | Listing of Important Protocol Deviations for Evaluable Subjects |
| 1.6 | | All Evaluable Subjects | Listing of Demographic Characteristics for Evaluable Subjects |
| 1.7 | | All Evaluable Subjects | Listing of Race Details |
| | 1.8 | All Evaluable Subjects | Listing of Specific Medical Conditions at Screening |
| | 1.9 | All Evaluable Subjects | Listing of Surgical/Diagnostic Procedures |
| 1.10 | | All Evaluable Subjects | Listing of Concomitant Medications |
| 1.11 | | All Evaluable Subjects | Listing of Relationship Between ATC Level 1, Ingredient, and Verbatim Text |
| 2.1 | | All Evaluable Subjects | Listing of IPSS |
| | 2.2 | All Evaluable Subjects | Listing of BPH-Related Health Status |
| 2.3 | | All Evaluable Subjects | Listing of BPE/BPO |
| | 3.1 | Screened But Not<br>Evaluable Subjects | Listing of All Adverse Events for Screened But Not Evaluable Subjects |
| 3.2 | | All Evaluable Subjects | Listing of All Adverse Events for Evaluable Subjects |
| 3.3 | | All Evaluable Subjects | Listing of Relationship Between System Organ Class and Verbatim Text |
| 3.4 | | All Evaluable Subjects | Listing of Subject Numbers for Specific Adverse Events |
| 3.5 | | All Evaluable Subjects | Listing of Fatal Adverse Events |
| 3.6 | | All Evaluable Subjects | Listing of Non-Fatal Serious Adverse Events |
| 3.7 | | All Evaluable Subjects | Listing of Adverse Events Leading to Withdrawal From the Study |
| 3.8 | | All Evaluable Subjects | Listing of Relationship Between Special Interest Adverse Events and Verbatim Text |
| 3.9 | | All Evaluable Subjects | Listing of Adverse Events of Special Interest |
| | 3.10 | All Evaluable Subjects | Listing of PSA (ng/mL) Values |
| | 3.11 | All Evaluable Subjects | Listing of Urine Dipstick and Urinalysis Data |
| | 3.12 | All Evaluable Subjects | Listing of Digital Rectal Examination Data |

# 11.16. Appendix 16: Example Mock Shells for Data Displays

Filed separately in IMMS.

# 11.17. Appendix 17: Amendment 01 Revision

| Item | RAP Revision General Description | RAP Section |
|---|---|---|
| 01 | Indicate RAP "Amendment Number 01" with administrative details including revision number, copyright year, effective date, description, author, and approver. | -Cover page -Document header -Section 1: Key Elements of the RAP -Section 2.1: Changes to the Protocol Defined Statistical Analysis Plan |
| 02 | Redefine the Analysis Populations as follows: Previous: Screened But Not Enrolled Population – Comprised of all subjects who are screened for eligibility but who do not meet the entry criteria. Current: Screened But Not Evaluable Population – Comprised of all subjects who are screened for eligibility, but do not qualify for the Evaluable Population. | -Section 1: Key Elements of the RAP -Analysis Populations -Section 4: Analysis Populations |
| | Previous: Enrolled Population - Comprised of all subjects who meet the entry criteria, including a positive IPSS screening result (score ≥8) and/or a positive BPE/BPO screening result (score ≥3). Current: Evaluable Population - Comprised of all subjects who meet the entry criteria, including a positive IPSS screening result (score ≥8) and/or a positive BPE/BPO screening result (score ≥3). Note: the population definition did not change for the | |
| 03 | Enrolled/Evaluable Population. Remove the following text: | -Section 6.2: Subject Accountability |
| | Number of subjects who were incorrectly enrolled with IPSS<8 and BPE/BPO<3. This bullet point is no longer needed in this section. This group of subjects will no longer need to appear on the Summary Table for Screened subjects since they will be included with the Number of Screened But Not Evaluable subjects. | Occion 6.2. Oubject Accountability |
| 04 | Update the names of the study populations as follows: Screened But Not Enrolled Population is changed to the Screened But Not Evaluable Population Enrolled Population is changed to the Evaluable Population. | -Section 4.1.1: Inclusion / Exclusion Criteria Deviations -Section 4.1.2: Important Protocol Deviations -Section 6.1: Overview of Planned Analyses -Table 2: Overview of Planned Study Population analyses |

| | | Cootion 6 2: Cubicat Assemble 11th |
|---|---|---|
| | | -Section 6.2: Subject Accountability -Section 6.3: Subject Disposition |
| | | -Section 6.4: Demographic |
| | | Characteristics |
| | | -Section 6.5: Medical Conditions, |
| | | Surgical procedures, and Concomitant |
| | | Medications |
| | | -Section 7.1.1: Overview of Planned |
| | | primary Efficacy Analyses |
| | | -Section 8.1.1 and Table 4: Overview of |
| | | Planned Secondary Efficacy Analyses |
| | | -Section 8.1.2.1: IPSS Screening Tool |
| | | -Section 8.1.2.3: BPE/BPO Screening |
| | | Tool |
| | | -Section 8.2.1: Overview of Planned |
| | | Analyses |
| | | -Section 8.2.2: Adverse Events |
| | | -Section 8.2.5: Clinical Laboratory |
| | | Assessments |
| | | -Section 8.2.6: Serum PSA |
| | | -Appendix 1: Protocol Deviation |
| | | Management and Definitions for Per |
| | | Protocol Population |
| | | -Section 11.1.1: Exclusions from Per |
| | | Protocol Population |
| | | -Appendix 6: Derived and Transformed |
| | | Data |
| | | -Section 11.6.1 General (Date of |
| | | Enrollment) |
| | | -Appendix 7: Premature Withdrawals |
| | | and Handling of Missing Data |
| | | -Section 11.7.1: Premature |
| | | Withdrawals |
| | | -Section 11.7.2 Handling of Missing |
| | | Data |
| | | -Appendix 15: List of Data Displays |
| | | -Section 11.15.2: Study Population |
| | | Tables |
| | | -Section 11.15.3: Efficacy Tables |
| | | -Section 11.15.4: Efficacy Figures |
| | | -Section 11.15.5: Safety Tables |
| | | -Section 11.15.6: ICH Listings |
| 05 | Revise title of Table 1.4 – Table 1.10, Table 1.14 – Table | -Appendix 15: List of Data Displays |
| | 1.17 | -Section 11.15.2: Study Population |
| | Daviss title of Figure 0.4. Figure 0.2 | Tables |
| | Revise title of Figure 2.1 – Figure 2.3 | -Section 11.15.4: Efficacy Figures |
| | Revise title of Listing 1.1 – Listing 1.2, Listing 1.5 – | -Section 11.15.6: ICH Listings |
| | 1.0.100 and of Elouing 1.1 Library 1.2, Library 1.0 | |

| Listing 1.6, Listing 3.1 – Listing 3.2 |
|---|
| Screened But Not Enrolled Population is changed to the Screened But Not Evaluable Population |
| Enrolled Population is changed to the Evaluable Population. |